# Clinical Intervention Study Protocol

# NCT03859076

FULL PROTOCOL TITLE Mindfulness-Based Blood Pressure Reduction: Stage 2a RCT

Study Chairman or Principal Investigator:
Eric B. Loucks, PhD
Associate Professor, Department of Epidemiology
Brown University School of Public Health

Supported by:
The National Center for Complementary and Integrative Health
5UH3AT009145-04

# Clinical Intervention Study Protocol

# **FULL PROTOCOL TITLE**

Mindfulness-Based Blood Pressure Reduction: Stage 2a RCT

# **Study Chairman or Principal Investigator:**

Eric B. Loucks, PhD
Associate Professor, Department of Epidemiology
Brown University School of Public Health

Supported by: The National Center for Complementary and Integrative Health

5UH3AT009145-04

**Study Intervention Provided by:** 

N/A

**Sponsor of IND (IDE):** 

N/A

## **Tool Revision History**

Version Number: 2.1 Version Date: July 6, 2018 Summary of Revisions Made:

- Revised sample size from 202 to 122. The total sample size of n=122 is comprised of n=50 for the MB-BP intervention group; n=50 for the enhanced usual care control group; and n=22 for the exploratory MBSR group. This sample size reflects recruitment during UH3 phase rather than during both the UH2 and UH3 phases.
- Mediation analyses will be performed via meta-analysis of both samples from the UH2 and UH3 phases, for which the participants were assessed using identical methods. This will maximize statistical power for mediation analyses, which require greater power.
- Narrowed primary outcome to one (Multidimensional Assessment of Interoceptive Awareness), in order to minimize issues of multiple statistical testing and maximize statistical power, given the smaller sample size when analyses are restricted to the data collected during the UH3 phase.
- A unique clinicaltrials.gov registration will be created based on the UH3-specific aims, data collection, and analyses.

Version Number: 2.2

Version Date: August 9th, 2018

Summary of Revisions Made: Replaced Dr. Wen-Chih Wu with Dr. Gaurav Choudhary as the clinical cardiologist on the DSMB. This was done because Dr. Wu and Dr. Loucks have published together in the past three year. Dr. Choudhary and Dr. Loucks have not published together.

Version Number: 2.3

Version Date: August 16, 2018 Summary of Revisions Made:

- Addressed comments and requested revisions per OCRA 8/9/18 review. Comments were relayed by Program Director, Merav Sabri, to study PI, Eric Loucks in an email sent on August 10, 2018.
- Revised Appendix B as requested by OCRA. Also removed sub-Appendix A, Conducting Orientation Sessions at the Center for Mindfulness in Medicine, Health Care and Society University of Massachusetts Medical School, as it is not utilized in this study
- Updated phone screener document (Appendix C) to reflect OCRA review comments and updated study protocol.
- Replaced informed consent form (Appendix D) with updated version (v.3.2)

Version Number: 2.4

Version Date: November 14, 2018

Summary of Revisions Made: The modifications made to the study protocol outlined below were largely the result of items brought to the research team's attention during the NCCIH/Westat September 13, 2018 Site Initiation Visit (SIV) and in the related SIV Report sent on October 9, 2018.

- Updated the study team roster to include the co-PI (King); data safety monitoring expert (Britton); and the study clinicians (Wu and Flynn).
- Clarified the role UMass Medical School will play in conducting the fMRI imaging study and explicitly stated that the details of said study will be documented separately.
- Removed the MBSR exploratory arm. (Refer to Nov. 6, 2018 PI email to NCCIH PO for rationale. NCCIH provided written approval in Nov. 12, 2018 email response to PI)
- Revised (clarified) descriptive language around recruitment; screening; inclusion criteria; blinding; randomization procedures; intervention timing, duration, and content; assessment windows; and data management to more accurately reflect the plan for UH3 study procedures.
- Updated the full list of measures for UH3, which included the removal of: actigraphy devices, Mindful Skill Acquisition scale, dietary self-efficacy, and the readiness to change for hypertenstive risk factors questionnaire. Additionally, the following measures were added: the PROMIS Global Health v.1.2 scale, childhood food insecurity questionnaire, alcohol consumption, mindfulness home practice questions, the Connor-Davidson Resilience scale, the Self-efficacy for chronic disease management questionnaire, and 6-month semi-structured exit interview questions.
- Revised Section 7 (Safety Assessments) to reflect the new Data safety and monitoring plan (DSMP) put forth for UH3.
- Clarified language around the estimated enrollment and analyzable sample size for the fMRI Study.
- Corrected clerical and grammatical errors and cleaned up the language to be more concise and clear.

Version Number: 2.5

Version Date: December 11, 2018

Summary of Revisions Made: Addressed the comments and requested clarifications sent to study PI (Loucks) by NCCIH Program Director (M. Sabri) on December 6, 2018 at 6:18 PM EST. The specific revisions include:

- Adding clarifying language on study randomization and cohort size to section 6.2.4 (Randomization and Intervention Allocation).
- Expounding upon circumstances that might possibly lead to Investigator-initiated withdrawals, which are discussed in section 7.3.3. of the Safety Assessment section of the protocol.

# TABLE OF CONTENTS

| | | | Page |
|---|---|---|---|
| C | linical In | tervention Study Protocol | 1 |
| F۱ | JLL PR | OTOCOL TITLE | 2 |
| | Tool Re | evision History | 3 |
| T | ABLE O | F CONTENTS | 5 |
| | MB-BP | STUDY TEAM ROSTER | 8 |
| | PARTIC | CIPATING STUDY SITES | 9 |
| | PROTO | DCOL SUMMARY | 9 |
| 1. | STUDY | OBJECTIVES | 12 |
| | 1.1 | Primary Objective | 12 |
| 2. | BACK | BROUND AND RATIONALE | 12 |
| | 2.1 | Background on Condition, Disease, or Other Primary Study Focus | 12 |
| | 2.2 | Study Rationale | 15 |
| 3. | STUDY | DESIGN | 15 |
| 4. | SELEC | TION AND ENROLLMENT OF PARTICIPANTS | 17 |
| | 4.1 | Inclusion Criteria | 17 |
| | 4.2 | Exclusion Criteria | 17 |
| | 4.3 | Study Enrollment Procedures | 17 |
| 5. | STUDY | 'INTERVENTIONS | 18 |
| | 5.1 | Interventions, Administration, and Duration | 18 |
| | 5.2 | Handling of Study Interventions | 19 |
| | 5.3 | Concomitant Interventions | 19 |
| | 5.4 | Adherence Assessment | 19 |
| 6. | STUDY | PROCEDURES | 21 |
| | 6.1 | Schedule of Evaluations | 21 |
| | 6.2 | Description of Evaluations | 22 |
| | 6.2.1 | Screening Evaluation and Consenting Procedure | 22 |
| | 6.2.2 | P. Enrollment | 22 |
| | 6.2.3 | Baseline Assessments | 22 |
| | 6.2.4 | Randomization and Intervention Allocation | 24 |

| | 6.2.5 | 5 Blinding | 25 |
|---|---|---|---|
| | 6.2.6 | 6 Follow-up Visits | 25 |
| | 6.2.7 | 7 Completion/Final Evaluation | 25 |
| 7. \$ | SAFET | TY ASSESSMENTS | 25 |
| - | 7.1 | Expected Risks and Specification of Safety Parameters | 25 |
| - | 7.2 | Methods and Timing for Assessing, Recording, and Analyzing Safety Parameters | 28 |
| - | 7.3 | Adverse Events and Serious Adverse Events, Reporting Procedures, and Follow-up | )28 |
| | 7.3.1 | 1 Mental Health | 29 |
| | 7.3.2 | 2 Physical Health | 30 |
| | 7.3.3 | 3 Other | 30 |
| - | 7.4 | Safety Monitoring | 31 |
| 8. I | NTER | VENTION DISCONTINUATION | 33 |
| 9. \$ | STATI | STICAL CONSIDERATIONS | 33 |
| ( | 9.1 | General Design | 33 |
| Ç | 9.2 | Sample Size and Randomization | 33 |
| Ç | 9.3 | Definition of Populations | 35 |
| Ç | 9.4 | Interim Analyses and Stopping Rules | 35 |
| Ç | 9.5 | Outcomes | 35 |
| | 9.5.1 | 1 Primary Outcome | 35 |
| | 9.5.2 | 2 Secondary Outcomes | 35 |
| ( | 9.6 | Data Analyses | 35 |
| 10. | DATA | A COLLECTION AND QUALITY ASSURANCE | 36 |
| | 10.1 | Data Collection Forms | 36 |
| | 10.2 | Data Management | 36 |
| | 10.3 | Quality Assurance | 36 |
| | 10.3 | 3.1 Training | 36 |
| | 10.3 | 3.2 Quality Control Committee | 36 |
| | 10.3 | 3.3 Metrics | 36 |
| | 10.3 | 8.4 Protocol Deviations | 38 |
| | 10.3 | 5.5 Monitoring | 38 |
| 11 | DADT | FICIDANT RIGHTS AND CONFIDENTIALITY | 38 |

| 11.1 I | Institutional Review Board (IRB) Review | 38 |
|-----------|----------------------------------------------------|----|
| 11.2 I | Informed Consent Forms | 38 |
| 11.3 F | Participant Confidentiality | 38 |
| 11.4 | Study Discontinuation | 38 |
| 12. COMM | MITTEES | 39 |
| 13. PUBLI | CATION OF RESEARCH FINDINGS | 39 |
| 14. REFE | RENCES | 39 |
| 15. SUPPI | LEMENTS/APPENDICES | 55 |
| Append | ix A MB-BP Curriculum Guide | 55 |
| Append | ix B MBSR Curriculum Guide | 55 |
| Append | ix C MB-BP Phone Screener (verbal consent process) | 55 |
| Append | ix D MB-BP Informed Consent | 55 |
| Append | ix E Anthropometric Quality Control Manual | 55 |
| Append | ix F Blood Pressure Quality Control Manual | 55 |

#### **MB-BP STUDY TEAM ROSTER**

Eric B. Loucks, Ph.D. Principal Investigator Brown University School of Public Health 121 South Main St., Providence, RI 02912

Phone: 401-863-6283 Fax: 401-863-3713

Email: eric.loucks@brown.edu

Jean A. King, Ph.D. Co-Principal Investigator 100 Institute Road, Worcester MA 01609-2280

Phone: 508-831-4677 Email: jaking@wpi.edu

Frances Saadeh, MPH Senior Project Coordinator 121 South Main St., Providence, RI 02912

Phone: 401-863-6361

Email: frances saadeh@brown.edu

Yu Li, PhD Statistician 121 South Main St., Providence, RI 02912 Phone: 401-863-6792

Phone: 401-863-6792 Email: yu\_li1@brown.edu

Roee Gutman, PhD Senior Statistician 121 South Main St., Providence, RI 02912

Phone: 401-863-2682

Email: rgutman@stat.brown.edu

#### **Study Clinicians**

Ellen Flynn, MD – Clinical Psychiatrist Women's Medicine Collaborative 146 West River Street, 3<sup>rd</sup> Floor, Providence, RI 02904 Phone: 401-793-7020

Email: eflynn@lifespan.org

Wen-Chih (Hank) Wu, MD, MPH – Cardiologist 164 Summit Ave, Providence, RI 02906 Providence, RI 02906

Phone: 401-793-5810 Fax: 401-793-5815

Email: wen-chih\_wu@brown.edu

#### **Data and Safety Monitoring Board (DSMB)**

Donald Edmondson, PhD, MPH DSMB Chair

622 W 168th Street, PH 9-317 New York, NY 10032

Phone: 212-342-3674 Fax: 212-305-0312

Email: dee2109@cumc.columbia.edu

Gaurav Choudhary, MD Providence VA Medical Center 830 Chalkstone Avenue Providence, RI 02908 Tel: 401-273-7100 ext 2029 Gaurav Choudhary@brown.edu

Tao Liu, PhD 121 South Main Street, Providence, RI 02912

Phone: 401-863-6480 Fax: 401-863-9182

Email: tliu@stat.brown.edu

#### **Data and Safety Monitoring Expert**

Willoughby Britton, Ph.D.
Director, Clinical and Affective Neuroscience Laboratory
Assistant Professor (Research)
Department of Psychiatry and Human Behavior
Warren Alpert Medical School at Brown University

Phone: 520-245-1855

Email: willoughby britton@brown.edu

#### **PARTICIPATING STUDY SITES**

There is one study site, Brown University, carrying out the Mindfulness-Based Blood Pressure Reduction (MB-BP) study protocol outlined in this document. The University of Massachusetts Medical School is conducting the fMRI Imaging study that will recruit and scan a subset of MB-BP study participants (see separate fMRI study protocol and related MOP for full detail).

#### PROTOCOL SUMMARY

#### **Study Title**

Mindfulness Based Blood Pressure Reduction: Stage 2a Randomized Controlled Trial

### **Objectives**

- 1. *Impacts of MB-BP on Primary Self-Regulation Targets:* Identify the impacts of MB-BP *vs.* enhanced usual care on the primary self-regulation target, specifically an assay of self-related processes (MAIA), described in Table 1. We hypothesize that MB-BP will significantly improve the MAIA in directions of better self-regulation, compared to control.
  - Secondary analyses will evaluate impacts on secondary self-regulation targets including an assay of emotion regulation (DERS), and cognitive processes (SART), described in Table 1.
  - b. Exploratory analyses will evaluate engagement of MB-BP vs. enhanced usual care with triangulated self-regulation target assays described in **Table 1** such as emotion regulation and stress (Pittsburgh Stress Battery, Perceived Stress Scale), self-related processes (Heart Beat Detection Task, Interoceptive Awareness fMRI Task), and cognitive processes (Mindful Attention Awareness Scale). Measures such as the neuroimaging Interoceptive Awareness fMRI Task will replicate assays in the MINDFUL-PC study.
- 2. Self-Regulation Targets as Mediators of MB-BP Effect on Medical Regimen Adherence and Health Behavior Change: Evaluate the degree to which the engagement of MB-BP with self-regulation targets translates into improved prehypertension/hypertension medical regimen adherence, specifically for the Dietary Approaches to Stop Hypertension (DASH)-consistent diet. We hypothesize that MB-BP will increase the DASH diet score compared to control, in participants with low DASH diet adherence at baseline (DASH diet score <5.5), and that the self-regulation primary outcome in Aim 1 (i.e. MAIA) is a significant mediator.</p>
- 3. Further develop an MB-BP therapist manual and training program, including procedures for training, supervising, and evaluating therapists. The PI will implement training he receives from the University of Bangor in the United Kingdom in May 2018 to implement the Mindfulness-Based Interventions Teacher Assessment Criteria (MBI-TAC) for MB-BP instructors, which is the most respected quantitative and qualitative tool developed to provide feedback for enhancing MBI teacher effectiveness, and establishing teacher certification.<sup>1-3</sup>

#### **Design and Outcomes**

During the UH3 phase, we will perform a Stage 2a<sup>4</sup> two-arm RCT of MB-BP vs. enhanced usual care control, enrolling 50 individuals aged 18 years of age and older per group. This is a pragmatic control group designed to inform physicians if MB-BP would be of service to refer patients, compared to enhanced usual care they could provide patients in well-resourced settings. This control group was decided upon through recommendations by the Research Coordinating Center at Columbia University, the Data Safety Monitoring Board, and several collaborating cardiologists and family physician clinician-researchers. Enhanced usual care involves every participant being provided with a validated home blood pressure monitor (Omron, Model PB786N), which has evidence in and of itself to potentially lower blood pressure. 5.6 and is beyond usual care at this time. All participants who have Stage 2 hypertension (blood pressure >140/90 mmHg) will be offered to have their physicians notified, if not already being overseen for uncontrolled hypertension. For participants with uncontrolled hypertension who do not have a physician, we will work with participants to provide access within constraints of their health insurance. Enhanced usual care group participants receive an educational brochure from the American Heart Association entitled "Understanding and Controlling Your High Blood Pressure Brochure" (product code 50-1731).

#### **Blinding**

All study staff will be blinded to the participant treatment allocation with the exception of the instructor, individual who performs the randomization, and staff member coordinating participants within each course. All staff performing participant assessments will be blinded to the participant treatment allocation to promote equipoise. Data analyses will be performed by a statistician blinded to treatment allocation type. The data manager will be able to break blinding if needed (e.g. for Data and Safety Monitoring Board).

#### Intervention Allocation

Stratified randomization will be used, as simple randomization can fail if it creates groups unbalanced for critical features known to affect outcomes.<sup>7,8</sup> Stratified randomization can reduce both types I and II error, improve trial efficiency, and facilitate subgroup and interim analyses.<sup>7</sup> Randomization will be done using an online computer software program known as Research Randomizer (Version 4.0).<sup>9</sup> The randomization process will occur after each new round of enrollment. Study enrollment will continue until target enrollment goals are reached (i.e., n=50 for MBBP intervention group, n=50 for enhanced usual care control group).

#### Interventions and Duration

Two-arm RCT comparing MB-BP vs. enhanced usual care. Follow-up assessments will take place within pre-defined assessment windows occurring around 10 weeks, 6 months, and 1 year post- intervention commencement. For participants on waitlist enhanced usual care, they will be offered MB-BP after the 6-month follow-up with no additional assessments unless they would like the assessments for follow-up information on changes in their health. Participants in the intervention group will be asked to come back at the 1-year follow up window for an abbreviated follow up assessment. Thus the total length of involvement for study participants will be up to one year from the time of enrollment to the time of the final research assessment. The study intervention lasts 9 weeks, may be nonconsecutive weeks in the event of a holiday or instructor availability, and takes place in the first three months for individuals in the intervention arm.

#### Sample Size and Population

We anticipate needing to recruit and enroll a total of 100 eligible individuals during Phase 3. This will consist of 50 individuals per group for both the MB-BP intervention arm and the enhanced usual care arm. (see Figure 1 below for detail).

For more detailed discussion of group allocation, stratification factors, and how it influences study population, please refer to Section 6.2.4.

#### Inclusion/exclusion criteria:

*Inclusion Criterion:* Elevated blood pressure defined as ≥120 mmHg systolic or ≥80 mmHg diastolic pressure; <sup>10</sup> able to speak, read, and write in English; all adults (≥18 years of age), genders and racial/ethnic groups are eligible to be included.

Exclusion Criteria: Exclusion criteria follow standard guidelines and recommendations:<sup>11</sup> (a) current regular meditation practice (>once/week); (b) serious medical illness precluding regular class attendance; (c) current substance abuse, suicidal ideation or eating disorder, (d) history of bipolar or psychotic disorders or self-injurious behaviors. These participants are excluded

because they may disrupt group participation, require additional or specialized treatment, or are already participating in practices similar to the intervention.

#### 1. STUDY OBJECTIVES

## 1.1 Primary Objective

- Impacts of MB-BP on Primary Self-Regulation Targets: Identify the impacts of MB-BP vs. enhanced usual care on the primary self-regulation target, specifically an assay of self-related processes (MAIA) described in Table 1. We hypothesize that MB-BP will significantly improve the MAIA in directions of better self-regulation, compared to control.
  - Secondary analyses will evaluate impacts on secondary self-regulation targets including an assay of emotion regulation (DERS), and cognitive processes (SART), described in Table 1.
  - b. Exploratory analyses will evaluate engagement of MB-BP vs. enhanced usual care with triangulated self-regulation target assays described in **Table 1** such as emotion regulation and stress (Pittsburgh Stress Battery, Perceived Stress Scale), self-related processes (Heart Beat Detection Task, Interoceptive Awareness fMRI Task), and cognitive processes (Mindful Attention Awareness Scale). Measures such as the neuroimaging Interoceptive Awareness fMRI Task will replicate assays in the MINDFUL-PC study.
- 2. Self-Regulation Targets as Mediators of MB-BP Effect on Medical Regimen Adherence and Health Behavior Change: Evaluate the degree to which the engagement of MB-BP with self-regulation targets translates into improved prehypertension/hypertension medical regimen adherence, specifically for the Dietary Approaches to Stop Hypertension (DASH)-consistent diet. We hypothesize that MB-BP will increase the DASH diet score compared to control, in participants with low DASH diet adherence at baseline (DASH diet score <5.5), and that the self-regulation primary outcomes in Aim 1 are significant mediators.
- 3. Further develop an MB-BP therapist manual and training program, including procedures for training, supervising, and evaluating therapists. The PI will implement training he receives from the University of Bangor in the United Kingdom in May 2018 to implement the Mindfulness-Based Interventions Teacher Assessment Criteria (MBI-TAC) for MB-BP instructors, which is the most respected quantitative and qualitative tool developed to provide feedback for enhancing MBI teacher effectiveness, and establishing teacher certification.<sup>1-3</sup>

#### 2. BACKGROUND AND RATIONALE

#### 2.1 Background on Condition, Disease, or Other Primary Study Focus

The World Health Organization reported that suboptimal blood pressure (BP) is responsible for more than half of cardiovascular disease mortality world-wide. Furthermore, greater than half of those with hypertension have uncontrolled BP.<sup>12</sup> <u>A 2009 Institute of Medicine report recommended prioritizing research to "Compare the effectiveness of mindfulness-based interventions (e.g. yoga, meditation, deep breathing training) and usual care in treating... cardiovascular risk factors." <sup>13</sup> Evidence-based mindfulness interventions, including Mindfulness-Based Stress Reduction, may have some effects on blood pressure, where a recent meta-analysis and systematic review of 4 randomized controlled trials demonstrated</u>

significant effects, but evidence of heterogeneity in effect sizes. <sup>14</sup> The methodologically highest quality studies had the smallest effect sizes (range 0-5 mmHg). <sup>14</sup> Mindfulness-Based Stress Reduction (MBSR) has been customized to a number of disease processes, such as Mindfulness-Based Cognitive Therapy for patients with recurrent depression, and Mindfulness-Based Relapse Prevention for patients with substance use addictions. <sup>15-17</sup> Effect sizes may be increased by customizing mindfulness interventions to diseases of interest. The same may be true for hypertension, *however mindfulness interventions customized for prehypertensive/hypertensive patients have never been investigated. Until methodologically rigorous studies to evaluate customized interventions for hypertension are performed, we will not know if the observed preliminary effects of general mindfulness interventions on blood pressure reduction could be much more effective with a tailored approach.* 

The development of effective interventions that enhance the capacity for self-regulation among people with chronic health conditions is a major public health challenge in the United States and worldwide. The process of healthcare system transformation that is underway focuses on moving accountability for healthcare costs to healthcare systems. 18 Meanwhile, in order to survive, healthcare systems must rapidly learn to deliver interventions that can enhance their patients' capacity to self-manage these deadly and costly chronic health conditions. 19 While access to care<sup>20</sup> and health education<sup>21</sup> are essential, a person's capacity for self-regulation is often the primary limiting factor in their ability to adhere to their medical regimen, collaborate on illness self-management, and reduce health risk behaviors. 22-25 Self-regulation refers to the process of managing cognitive, emotional, and self-relevant resources to align mental states and behavior with goals.<sup>26-28</sup> Changing risk behaviors that influence hypertension risk, such as physical inactivity, diet, excessive alcohol use, and poor medication adherence, requires skills for self-regulation that are broadly applicable within multiple environments. A research collaboration that could test methods for engaging self-regulation mechanisms, identify specific target tests, and rapidly integrate these into an empirically-optimized clinical interventions that are ready for implementation and rapid dissemination within health care settings for patients with chronic illness would make a substantial impact on chronic illness management and the entire healthcare system. Mindfulness-Based Interventions (MBIs) have already begun to offer feasible basic building blocks for the rapid integration of an empirically-optimized, transdiagnostic, self-regulation toolkit into healthcare across multiple contexts and age groups.

Mindfulness meditation, a form of training that involves maintaining a non-judgmental form of attention to immediate experience, <sup>29</sup> has been employed in both clinical and non-clinical settings to facilitate self-regulation and behavior change. <sup>30-34</sup> Mindfulness-Based Interventions (MBIs), <sup>35</sup> sometimes referred to as "3<sup>rd</sup> Wave Behavioral Therapies," <sup>36</sup> have become widely used in both clinical and non-clinical settings, including prisons, <sup>37,38</sup> the military, <sup>39-41</sup> and both K-12<sup>42-45</sup> and higher education, <sup>46</sup> and are emerging as a wide-spread, potentially cost-saving, <sup>47</sup> comprehensive methods for enhancing self-regulation in multiple medical contexts. *While MBIs efficacy has been demonstrated for several conditions related to self-regulation,* <sup>48-50</sup> the field lacks consensus about the mechanisms through which these interventions engage self-regulatory processes and impact of MBIs on medical regimen adherence and health behavior changes. Without this knowledge, a plethora of MBIs are being developed without systematically building on discoveries of which components of the interventions have the most impact on specific health behaviors and outcomes. As a result, the interventions are not as rigorous in their design, which may limit their efficacy and account for some of the mixed results found in the literature.

Self-regulation requires both *initiating* behavior change and *maintaining* behavior change,<sup>51,52</sup> implying corrective adjustments originating within a person and taking place as needed in order

to maintain and sustain the intended goal. Self-regulatory failure is primarily determined by deficits in (or depletion of) self-regulatory strength, <sup>53</sup> highlighting the need for interventions that strengthen self-regulation capacity. Current behavioral models lack a full integration of tools for strengthening self-regulation towards both initiation and maintenance of behavior change. 51,52 Strategies focusing on extrinsic rewards or behavioral economics can help change behavior, but intrinsic motivation is ultimately essential to self-regulation.<sup>54</sup> Behavioral and psychological therapies can provide emotional regulation strategies and some even include motivational components: 55,56 however, they generally lack tools to strengthen core cognitive resources, such as attention and inhibitory control, which are necessary to support maintenance of behavior change. In contrast, MBIs uniquely integrate training in the emotional, motivational, and cognitive aspects of self-regulation within one therapeutic intervention. By frequently returning attention to the present moment with a specific orientation to experience (curious, open-minded, and accepting), mindfulness practice strengthens the capacity for frequent daily corrective adjustments needed to stay on track with intended goals. Studying how common self-regulation targets influence, and are influenced by, various components of MBIs provides a unique opportunity to develop an easy-to-disseminate, integrated therapeutic intervention optimized with the most potent components for enhancing self-regulation within the context of medical regimen adherence and the initiation and maintenance of health behaviors.

Following recent proposals on the mechanisms of action of mindfulness by our group<sup>30,57</sup> and others, <sup>58-62</sup> three broad self-regulation domains of mindfulness can be identified:

- (A) Cognitive processes, including attention (i.e. orienting, alerting, 63,64 vigilance, 65 and conversely sleepiness, cognitive fatigue, attentional lapses, and mind-wandering 66); executive function, conflict monitoring, 67,68 impulsivity and inhibitory control, 69,70 and metacognitive awareness. 71-73 Many studies indicate that meditation training, such as MBIs, engage these cognitive processes. 74-87
- (*B*) *Emotion regulation*, which is the capacity to alter the magnitude or duration of an emotional response.<sup>88</sup> Poor emotion regulation impairs the capacity for self-regulation behaviors that support health behaviors<sup>89-92</sup>, including medical regimen adherence.<sup>93</sup> MBIs favorably engage measures of emotion regulation such as amygdala activation,<sup>79,94-97</sup> sympathetic hyperarousal,<sup>98-103</sup> and emotional responses to stressful situations,<sup>102,104-111</sup> although opposite findings have also been reported<sup>112-114</sup> which leads to the question (to be addressed by this collaborative) of which conditions affect target engagement.
- (C) Self-related processes, including: (i) self-efficacy the belief in one's capabilities to execute the courses of action required to manage prospective situations (such as changing and maintaining a medical regimen), 115,116 which is a central aspect of self-regulation and changes in health behavior; 117,118 (ii) self-compassion the capacity to extend compassion to oneself in instances of perceived inadequacy or failure rather than engaging in either self-destructive behaviors (self-judgment, isolation, rumination) or in permissive, risky behaviors: 119-121 self-compassion has been found to promote health behaviors such as adhering to diets, 122 smoking cessation, 123 physical activity, 124 and seeking medical treatment when needed; 125 (iii) self-related rumination or mind-wandering which may be beneficial in some cases 126-128 but detrimental in others 129-133 and is a central topic in MBI research, by our group 57,134 and others; 135 and (iv) interoceptive awareness the awareness of internal manifestations of emotions and feelings, considered fundamental to the 'experiencing self', 136-141 a particular form of awareness which can be enhanced by the paying of purposeful, nonjudgmental attention ('mindfulness') to inner body sensations, 32,33,142 which is also of major interest in MBI research. 30,62,135,143-160

Consequently, we propose to conduct a Stage 2a behavioral intervention study to evaluate whether MBSR customized to pre-hypertensive and hypertensive patients has the potential to provide clinically relevant reductions in BP.

#### 2.2 Study Rationale

The MB-BP Study aims to customize the standardized MBSR¹6¹-¹6⁴ intervention to adult participants with prehypertension or uncontrolled hypertension. Similar to MBSR, the MB-BP intervention consists of eight 2.5-hour weekly group sessions (plus a 2.5-hour orientation session) and an 8-hour one-day session, led by a certified MBSR instructor with extensive cardiovascular disease and hypertension expertise.¹65-178 MB-BP builds a foundation of mindfulness skills (e.g. meditation, self-awareness, etc.) through the MBSR curriculum. MB-BP then directs attention towards hypertension risk factors. The unique areas of MB-BP are education on hypertension risk factors, hypertension health effects, and specific mindfulness modules focused on awareness of diet, physical activity, medication adherence, weight loss, and alcohol consumption and their effects on well-being. A curriculum guide has been created based on the standardized MBSR manual (**Appendix A**), and was further developed through the approaches described above, and sequentially revised based on participant feedback and preliminary findings.¹63,164 MB-BP participants learn a range of mindfulness skills including body scan exercises, meditation and yoga. Homework consists of practicing skills for ≥45 min/day, 6 days/week.

#### 3. STUDY DESIGN

We will perform a Stage 2a<sup>4</sup> two-arm RCT of MB-BP *vs.* enhanced usual care control. This is a pragmatic control group designed to inform physicians in well-resourced settings if MB-BP would be of service to refer patients to as compared to enhanced usual care patients. The study is intended to evaluate the impacts of MB-BP on the primary self-regulation outcome of interoceptive awareness (i.e. MAIA) as compared to an enhanced usual care group. Secondary self-regulation outcomes are described in the Objectives section outlined previously. This study also aims to evaluate the degree to which the engagement of MB-BP with self-regulation targets translates into improved prehypertension/hypertension medical regimen adherence, specifically for the Dietary Approaches to Stop Hypertension (DASH)-consistent diet.

The enhanced usual care control group was decided upon through recommendations by the Research Coordinating Center at Columbia University, the Data Safety Monitoring Board, and several collaborating cardiologists and family physician clinician-researchers. Enhanced usual care involves every participant being provided with a validated home blood pressure monitor (Omron, Model PB786N),<sup>179</sup> which has evidence in and of itself to potentially lower blood pressure, and is beyond usual care at this time.<sup>6,180</sup> All participants who have Stage 2 hypertension (blood pressure >140/90 mmHg) will be offered to have their physicians notified, if not already being overseen for uncontrolled hypertension. For participants with uncontrolled hypertension who do not have a physician, we will work with participants to provide access within constraints of their health insurance. Enhanced usual care group participants receive an educational brochure from the American Heart Association entitled "Understanding and Controlling Your High Blood Pressure Brochure" (product code 50-1731).

All research assessments will take place in the Brown University Mindfulness and Cardiovascular Health Lab in Providence, RI. The MB-BP intervention classes will be offered in both a University and community-based setting.

Baseline assessments for all enrolled participants will take place within four weeks of the start of the intervention. Follow-up assessments will take place during the 10 week, 6 month, and 1 year assessment windows, which are defined as: (a) "10 week" follow up assessments are to occur at least one day after and up to five weeks after the end of the intervention (i.e. the Week 8 class). Staff will prioritize completing the assessments within the first three weeks of the assessment window, but will allow for participants to complete up to five weeks after. (b) The "6-month" follow up assessments will be scheduled to occur six months from the orientation class date plus or minus 2.5 weeks. This allows for a five-week data collection period with prioritization given to the three-week window surrounding the official six-month date. (c) The "1 year" follow up assessments are to be completed with the intervention group participants only and will occur one year plus or minus a month after the start of the intervention (i.e., orientation date).

If a participant is unable to complete an assessment within the defined data collection window, but still wishes to participate, we will allow for the participant to complete an online home survey and/or in person follow up assessment beyond the parameters defined above.

Participants who were randomized to the waitlist enhanced usual care group will be offered MB-BP after the 6 month follow-up assessment is complete with no additional assessments unless they would like the final one year assessment for follow-up information on

Figure 1. Sampling approach and estimated participation rates for UH3 phase 3, consistent with CONSORT guidelines Not meeting inclusion criteria (n=39) Decline to participate (n=16) Allocated to enhance usual care control (n=50) to participate Excluded (n=55) Lost to follow-up Analyzed (n=44) Assessed for eligibility (n=155) ited intervention (n=45) allocated intervention Allocated to MBBP intervention (n=50) Receive allocated intervention Do not receive allocated intervention (n=5)Lost to follow-up (n=6) Discontinue interventio Analyzed (n=44) Enrolment Analysis Follow-up Allocation

changes in their health. Thus the total length of involvement for study participants will be up to one year from the time of enrollment to the time of the final research assessment. The study intervention lasts 9 weeks and takes place in the first two months for individuals in the intervention arm. The intervention will be offered several times a year over the course of the total study duration.

Prehypertension/Hypertension Medical Regimen Adherence Outcomes Assessment Methods:

Primary Prehypertension/Hypertension Medical Regimen Adherence Outcome: Dietary Approaches to Stop Hypertension (DASH) eating pattern score, <sup>181</sup> measured via 80-item Willet food frequency questionnaire, <sup>182</sup> assessing adherence to American Heart Association/American College of Cardiology (AHA/ACC) clinical practice hypertension guidelines DASH eating pattern score (range 0-8). <sup>10,181,183</sup>

Secondary outcomes of medical regimen adherence include the following: (1) Alcohol consumption: Amount and frequency of alcohol consumption, will be assessed via self-report utilizing standard questions from the Behavioral Risk Factor Surveillance Survey.¹84 AHA/ACC hypertension clinical practice guideline cut-point of healthy alcohol intake is ≤ 2 drinks (e.g. 24

oz. beer, 10 oz. wine, or 3 oz. 80-proof whiskey) per day in men and ≤1 drink per day in women. (2) Electronically-Measured Antihypertensive Medication Adherence: measured continuously using electronic medication bottle caps (eCAPS, Ottawa, Canada) Body Mass Index: height and weight directly assessed using standard epidemiologic methods, with change evaluated in participants considered overweight or obese (BMI≥25 kg/m²). (4) Physical activity: measured using the International Physical Activity Questionnaire which has undergone substantial validity and reliability testing. Adherence to Joint National Commission-7 (JNC-7) guidelines is 30 min aerobic physical activity ≥4 days per week.

Please see Section 6.2.4 for randomization, blinding and stratification methods.

Please see **Figure 1** for study groups including sample sizes. Please note that sample size recruited for the UH3 phase will be 50 participants per group for MB-BP and enhanced usual care control.

#### 4. SELECTION AND ENROLLMENT OF PARTICIPANTS

#### 4.1 Inclusion Criteria

Elevated blood pressure or hypertension defined as ≥120 mmHg systolic or ≥80 mmHg diastolic pressure. 10 Able to speak, read, and write in English. All adults (≥18 years of age), genders and racial/ethnic groups are eligible to be included.

#### 4.2 Exclusion Criteria

Exclusion criteria follow standard guidelines and recommendations:<sup>11</sup> (a) current regular mindfulness meditation practice (>once/week); (b) serious medical illness or cognitive condition (e.g., dementia) precluding regular class attendance and/or participation; (c) current substance abuse, suicidal ideation or eating disorder, (d) history of bipolar or psychotic disorders or self-injurious behaviors. These participants are excluded because they may disrupt group participation, require additional or specialized treatment, or are already participating in practices similar to the intervention. Additionally, we will be asking participants randomized to the control group to restrain from engaging in any type of formal mindfulness practice more than weekly during the first six months of study involvement so as to not introduce confounding variables. Individuals will be made aware of this requirement at the time of informed consent (first in-person screening). Anyone who is unwilling to follow the treatement requirement would be ineligible for the study.

#### 4.3 Study Enrollment Procedures

Participants will be recruited in part through cardiology and family practices via established relationships with physicians in Rhode Island and Massachusetts. Graduates from the MP-BP program have proven effective at recruiting their contacts. Furthermore, advertisements will be posted throughout Rhode Island and southern Massachusetts, and distributed via social media, inviting participants interested in lowering their blood pressure to enroll. Additionally, we will partner with local providers to recruit hypertensive patients through methods such as direct mailings and targeted recruitment at the Rhode Island Hospital Emergency Department.

Participants are randomly assigned a participant identifier at the time of screening. The key to participant name and identifier is kept in a secure location separate from the research data. The outcome of every screener completed is recorded in a password protected tracking system and reason for ineligibility is noted. Circumstances surrounding situations where eligible participants decline participation and cases where participants enroll but later withdraw are also documented in a tracking system.

Informed consent is collected at the time of the first in-person screener. Individuals wishing to enroll in the study are provided two copies of the written informed consent form which has been approved by the Brown University Institutional Review Board (IRB). In addition to allowing the participant time to read over the consent form, trained research staff review the important points of consent with each participant. The informed consent process is documented. A signed copy of the consent is kept on file in a secure location in the research lab separate from study data and a copy is offered to the participant to keep with his/her personal records. Due to the nature and delivery of the intervention, all participants must be able to read and write in English and be able to provide informed consent for their participation.

#### 5. STUDY INTERVENTIONS

#### 5.1 Interventions, Administration, and Duration

MB-BP Intervention Description: This study proposes to customize MBSR to participants with prehypertension/hypertension creating an intervention called Mindfulness Based Blood Pressure Reduction Study (MB-BP). Specifically, MB-BP is based on the standardized MBSR intervention described elsewhere, 161-164 and will consist of eight 2.5-hour weekly group sessions, a 2.5 hour orientation, and an 8hour one-day session. MB-BP will be performed by qualified or certified MBSR instructors<sup>190</sup> with formal training in cardiovascular health (e.g. dietician, physician assistant, health and wellness coach, and those with an Associate's or Bachelor's degree in relevant health sciences), and further certification in MB-BP, MB-BP instructor training involves: (1) An initial 40 hour in-person or online videoconference training where the unique elements of MB-BP are introduced. (2) Two half-day inperson training retreats where MB-BP-specific teaching modules are practiced in peer groups, supervised by the senior MB-BP trainer, with peer and trainer feedback. (3) Studying specific evidence-based articles on hypertension etiology, treatment and prevention, as well as articles synthesizing evidence of mindfulness on hypertension and hypertension risk factors. 10,183,191-193 A written exam evaluates knowledge in this area, for which instructors-in-training need to pass. (4) Supervised teaching of MB-BP in non-study participants is done using the Mindfulness-Based Intervention Teacher Assessment Criteria (MBI-TAC), 1,2,194 and an annotated MB-BP Curriculum Guide until adequate quality is established within predefined criteria.

The unique areas of MB-BP are education on hypertension risk factors, hypertension health effects, and specific mindfulness modules focused on awareness of diet, physical activity, medication adherence, alcohol consumption, stress, and social support for behavior change. A Curriculum Guide has been created based on the standardized MBSR manual developed at UMass Medical School (**Appendix B**). 163,164 MB-BP sessions contain instruction and practice in mindfulness meditation, and conversations about stress and coping. Students learn a range of mindfulness skills including body scan exercises, meditation and yoga. Homework consists of

practicing skills for ≥45 min/day, 6 days/week. All MB-BP classes are to be held in either University or community-based locations in a comfortable, accessible environment where privacy is able to be maintained.

MB-BP builds a foundation of mindfulness skills (e.g. meditation, self-awareness, etc.) through the MBSR curriculum. MB-BP then directs attention towards hypertension risk factors. Early in the MB-BP, the importance of hypertension for health and mortality is described, along with hypertension risk factors. Participants will have their blood pressure and hypertension risk factors assessed at baseline. and be provided with this information during the first in-person MB-BP session. This phase aims to engage participants' interest in hypertension risk factors, and increase motivation for behavior change. MB-BP encourages participants to explore personal readiness for change in the different hypertension risk factors, and explore utilizing mindfulness practices to engage with those risk factors that they choose to. Each week, focus is provided on different hypertension risk factors. However, common themes exist across all hypertension risk factors including (1) awareness of thoughts, emotions and physical sensations particularly surrounding hypertension risk factors such as overconsumption of palatable foods, sedentary activities, alcohol consumption, medication adherence; (2) craving, particularly for hypertension risk factors such as overconsumption of palatable foods, sedentary activities, and alcohol consumption; (3) the impact of bringing mindfulness to every moment, particularly in relation to hypertension risk factors. For example, when consuming highly palatable food, bringing awareness to the emotions, thoughts and physical sensations prior to eating, during eating, and in the time afterwards. Participants are trained to bring non-judgmental attention to the often short-term pleasure of overconsumption of foods, sedentary activities, heavy alcohol consumption, or not taking medications, and bring non-judgmental attention to the longer term suffering associations with these activities. Through this process, participants are encouraged to reflect on if behavioral choices provide more benefit or harm to their well-being, and to choose the behaviors that bring benefit. (4) Self-care: as awareness of thoughts, emotions and physical sensations increases, and self-regulation will likely increases as a result of the meditation practices, the curriculum will emphasize to participants that it is common for people to start caring for themselves more. It is a way of better knowing ourselves, and through knowing ourselves in in each moment, we often want to care for ourselves in each moment. This may mean taking medication that will help our health, or being more physical active, eating more healthily, or consuming more moderate amounts of alcohol.

#### 5.2 Handling of Study Interventions

Please see Appendices A and B for the MBSR and MB-BP curriculum guides.

#### 5.3 Concomitant Interventions

Please see inclusion/exclusion criteria in Sections 4.1 and 4.2.

#### 5.4 Adherence Assessment

Adherence to the prescribed MB-BP practices will be monitored through class attendance, practice logs and weekly health goals. Adherence data will be collected weekly during the course of the intervention. Dr. Schuman-Olivier is testing more

technologically enhanced forms of meditation logs (e.g. accelerometer-based ecological momentary assessment and actigraphy score; NCT01314378), and found large proportions of participants had difficulty using the device properly (e.g. failing to stop meditation timers), which hampered data quality (*paper in progress*). We discussed this issue with leading meditation researchers, and meditation logs remain their recommended method at this time. However, innovative approaches are being explored by Dr. Lazar, including smartphone apps linked to audio homework files, with timers linked to data exports. These technologies are not yet ready for use, but we will incorporate technological advances for homework monitoring once demonstrated to be effective. Data analyses will evaluate effect modification by adherence to the MB-BP practices.

## **6. STUDY PROCEDURES**

#### 6.1 Schedule of Evaluations

| | Assessment Times | | | |
|---|---|---|---|---|
| Variables Measured | Baseline | 10 weeks | 6 months | 1 year* |
| Demographics | Х | | | |
| Family history of hypertension | X | | | |
| Childhood Socioeconomic Status | X | | | |
| Adverse Childhood Experiences | X | | | |
| Depressive Symptomatology | X | X | X | |
| Anxiety | X | X | X | |
| Medication Use | X | X | X | X |
| Anti-Hypertensive Medication Adherence | X | X | X | |
| Blood pressure | X | X | X | X |
| Anthropometry | X | X | X | X |
| Physical Activity | X | X | X | |
| Diet | X | X | X | X |
| Alcohol consumption | X | X | X | X |
| Cigarette Smoking | X | X | X | |
| Sleep Duration | X | X | X | X |
| Mindfulness | X | X | X | |
| Mindfulness home practice | X | X | X | X |
| Emotional Eating | X | X | X | |
| Self-Compassion | X | X | X | |
| Perceived Stress | X | X | X | |
| Emotional Regulation | X | X | X | X |
| Interoception | X | X | X | X |
| Heartbeat Detection | X | X | X | |
| Decentering | X | X | X | |
| Attention Control | X | X | X | |
| Craving for Hypertensive Risk Factors | X | X | X | |
| Social Integration | X | X | X | |
| Loneliness | X | X | X | |
| PROMIS Global Health | X | X | X | |
| Self-Control | X | X | X | |
| Resilience | X | X | X | |
| Self-efficacy for managing chronic disease | X | Χ | Χ | |
| Stress Reactivity | X | X | X | |
| Delay Discounting | X | Χ | Χ | |
| Semi-structured exit interviews at 6 months | | | X | |

<sup>\*1-</sup>year assessments consist of a subset of the other two follow ups and will be completed only with intervention group as controls are offered course post 6-month follow-up

#### 6.2 Description of Evaluations

#### 6.2.1 Screening Evaluation and Consenting Procedure

Please see **Appendices C and D** for the consenting process prior to the phone screening, and prior to the in-person screening.

Final screening evaluations will occur at least one week prior to baseline assessments. Baseline assessments will occur within 4 weeks of intervention initiation.

Phone-Based Screening: For people who indicate interest in the study, this screening will take place by phone using trained research assistants to assess the exclusion criteria described above, with the exception of blood pressure which will be assessed in-person

*In-Person Screening:* If participants remain eligible after the phone-based screening, they will attend an in-person screening for blood pressure and medication assessment. If mean blood pressure is elevated (≥120 mmHg systolic and/or ≥80 mmHg diastolic pressure), participants will be invited to return for a second blood pressure reading. At that time, if the mean blood pressure across both assessment times is ≥120 mmHg systolic or ≥80 mmHg diastolic pressure, they will be invited to participate in the study.

#### 6.2.2 Enrollment

The enrollment date is the day that the individual has met all the screening criteria, signs the informed consent form, and confirms agreement to participate in the study.

#### 6.2.3 Baseline Assessments

- (1) Demographics: age, race/ethnicity, socioeconomic status (education, employment), and household structure.
- (2) Family History of Hypertension (FH): Assesses biological parents' history of having hypertension, based on questions from New England Family Study LEAP Project.
- (3) Childhood socioecononomic status: retrospective reporting of parents' education, based on standardized questionnaires used in the Atherosclerosis Risk in Communities (ARIC) study.
- (4) Adverse Childhood Experiences: Measured using the standardized Childhood Trauma Questionnaire (CTQ), Childhood food insecurity questionnaire, and the Childhood Experiences of Care and Abuse Inventory neglect subscale. 184,195-200
- (5) Depressive symptomatology: Assessed using Center for Epidemiologic Studies Depression Scale Revised (CESD-R). The CESD survey has been used extensively in the epidemiologic literature to assess depressive symptomatology.<sup>201</sup> The scale was updated to the CESD-R by Van Dam *et al.*, which allows diagnosable criteria similar to Diagnostic and Statistical Manual (DSM) of Mental Disorders.<sup>202</sup>
- (6) Anxiety: Assessed using the validated Beck Anxiety Inventory. 203-209
- (7) Medication use: Assessed directly from participants' medication bottles and selfreport using standardized forms, including medication name, dose, frequency of use, and reason of use.
- (8) Antihypertensive medication adherence: measured continuously using electronic medication bottle caps (eCAPS, Ottawa, Canada).<sup>185</sup>

- (9) Systolic and diastolic blood pressure: Clinical blood pressure will be measured using a calibrated Omron HEM-705CPN following American Heart Association and Joint National Committee (JNC) guidelines. 183,210,211 Additionally, participants will be asked to complete three at home blood pressure readings using a validated home blood pressure monitor (Omron, Model PB786N) provided at baseline.
- (10) Anthropometry: height and weight directly assessed using standard epidemiologic methods.<sup>186</sup>
- (11) Physical activity: The International Physical Activity Questionnaire which has undergone substantial validity and reliability testing. 187-189 Adherence to Joint National Commission-7 (JNC-7) guidelines is 30 min aerobic physical activity ≥4 days per week. 183
- (12) Diet: assessed utilizing the validated Food Frequency that allows for calculation of hypertension-related dietary factors, including salt intake, alcohol consumption, total caloric consumption, fruit and vegetable consumption, and Dietary Approaches to Stop Hypertension (DASH) eating pattern score.<sup>182</sup>
- (13) Alcohol consumption: additional self-report standardized questions assessing current alcohol consumption taken from the Behavioral Risk Factor Surveillance Survey (BRFSS).<sup>212</sup>
- (14) Cigarette smoking: current smoking assessed using self-report standardized questions from the New England Family Study.
- (15) Sleep duration: Sleep duration is assessed using a single question on sleep duration from the validated Pittsburgh Sleep Quality Index (PSQI).<sup>213-215</sup>
- (16) Mindfulness: Assessed using the validated Five Facet Mindfulness Questionnaire.<sup>216</sup>
- (17) Mindfulness Home Practice: questions capturing individuals at home mindfulness practice pre- and post- intervention are administered at each of the time points.
- (18) Emotional eating: measured using the Three Factor Eating Questionnaire Revised 21-item (TFEQ-R21).<sup>217,218</sup>
- (19) Self-compassion: Assessed using the validated Self-Compassion Scale Short Form (SCS-SF). 121
- (20) Perceived stress: Assessed using the validated 14-item Perceived Stress Scale. 219,220
- (21) Emotion regulation: Measured using the validated Difficulties in Emotion Regulation Scale.<sup>221</sup>
- (22) Interoception: Assessed directly using the Heartbeat Detection Task and in secondary self-report using the validated Multidimensional Assessment of Interoceptive Awareness (MAIA).<sup>222-225</sup>
- (23) Decentering: Assessed using the validated Experiences Questionnaire. 226,227
- (24) Attention control: Assessed using the Sustained Attention to Response Task (SART). The SART is a validated computerized test of sustained attention, response inhibition (executive function) and self-regulation.<sup>228-230</sup> <sup>231-233</sup>
- (25) Craving: craving for hypertension risk factors, including palatable foods, alcohol, and sedentary activities will be assessed using the validated Craving Experiences Questionnaire. <sup>234</sup>
- (26) Social integration: Measured using the validated 12-item Interpersonal Support Evaluation List (ISEL-12) measure of social support.<sup>235</sup>
- (27) Loneliness: Assessed using the validated R-UCLA Loneliness Scale. 236
- (28) Global Health: individual physical, mental and social health are measured using the validated NIH PROMIS Global Health v1.2 scale.<sup>237</sup>

- (29) Self-control: assessed using the validated Self-Control Scale short form. 238,239
- (30) Resilience: measured using the validated 10-item Connor-Davidson Resilience Scale (CD-RISC-10).<sup>240</sup>
- (31) Self-efficacy for chronic disease management: measured using the 6-item Self-efficacy for Managing Chronic Disease scale (SECD-6).<sup>241</sup>
- (32) Stress Reactivity: Assessed using the Pittsburg Stress Battery a standardized protocol of 3 computerized tasks designed to induce a stress response indicated by evaluated cardiovascular (CV) reactivity.<sup>242</sup>
- (33) Delayed Discounting: Assessed using the validated 5-Trial Adjusting Delay Discounting Task. <sup>243</sup>
- (34) Functional Magnetic Resonance Imaging (fMRI): Participants in the UH3 phase who elect to take part in the fMRI imaging study will undergo an fMRI scanning session for approximately 40 minutes at baseline and 10-week follow-up. Scans will be acquired with a 3T scanner while the subject is in the resting state. Final sample size will be 24 per group (n=48); enrolling up to 60 participants in total to reach target sample size. Participants will undergo a separate informed consent and screening process for the fMRI imaging, so that they can be in the MB-BP study without imaging if they prefer. Refer to the separate fMRI study protocol for details.

#### 6.2.4 Randomization and Intervention Allocation

Randomization will occur following the completion of baseline assessments prior to the initiation of study intervention. Only individuals who complete the baseline assessments and indicate they are available for the upcoming courses will be included in the randomization process.

Stratified randomization will be used, as simple randomization can fail if it creates groups unbalanced for critical features known to affect outcomes.<sup>7,8</sup> Stratified randomization can reduce both types I and II error, improve trial efficiency, and facilitate subgroup and interim analyses. 7 Variables used to create strata include age (≤60 vs. >60 years), gender (male vs. female), and/or uncontrolled hypertension (≥140 mmHg systolic pressure, or ≥90 mmHg diastolic pressure) vs. prehypertension (120 to <140 mmHg systolic pressure, and 80 to <90 mmHg diastolic pressure). Simple random sampling will occur within each of the eight strata, thus allowing for each arm of the study to be more balanced with respect to age, gender, and hypertension category. The total size of each stratum will vary from cohort to cohort. To conduct the randomization, a list of participant IDs and strata characteristics will be provided, and a trained researcher not affiliated with the study will perform the randomization on participants after baseline assessment and final determination of eligibility is complete. Randomization will be done using an online computer software program known as Research Randomizer (Version 4.0).9 The randomization process will occur after each new round of enrollment (i.e., unique cohort). If the cohort sample size is such that there are not enough participants for balance within the three strata, we will prioritize stratification by two key strata instead of three, specifically by baseline blood pressure status and gender. Furthermore, after randomization within strata, if sample sizes in the entire sample for cohort differ by more than one participant per group, then all imbalanced groups are re-randomized until the entire sample differs by no more than 1 participant per group (e.g. n=8 MB-BP, n=9 enhanced usual care control). Expected cohort sizes, consistent with the

SARP are 15-20 participants. We anticipate needing to run 6 to 7 cohorts to reach the target sample size.

Study enrollment will continue until target enrollment goals are reached (i.e., n=50 for MBBP intervention group and n=50 for enhanced usual care control group).

#### 6.2.5 Blinding

All study staff will be blinded to the participant treatment allocation with the exception of the instructor, individual who performs the randomization, and staff member coordinating participants within each course. All staff performing participant assessments will be blinded to the participant treatment allocation to promote equipoise. Data analyses will be performed by a statistician blinded to treatment allocation type. The data manager will be able to break blinding if needed (e.g. for Data and Safety Monitoring Board). Circumstances for breaking the blind would be a large number of adverse experiences (>10% of enrolled participants reporting AEs rated as severe or life threatening) taking place in one or more study group. In this case, the data safety monitoring board would be notified, and could break the blind to help determine the cause of the adverse experiences.

#### 6.2.6 Follow-up Visits

Follow-up assessments will be scheduled and conducted within the pre-defined assessment windows outlined previously in section 3, study design. Questionnaires and assessments administered at 10 weeks and 6-months follow-up are identical to those administered at the first in-person screening assessment and at baseline, with the exception that questionnaires for which the answers should not change or be informative (age, race/ethnicity, education, adverse childhood experiences, family history of hypertension) are not given at follow-ups. In addition, adverse events are monitored and documented at each of the follow-up periods as well as throughout the duration of an individual's study involvement according to the data safety monitoring protocol put forth in this grant. Participants are also asked a set of semi-structured questions at the end of their six month follow up that inquire about their experience as either a control group member or intervention group participant.

#### 6.2.7 Completion/Final Evaluation

For control group participants, the 6-month evaluation is the final visit. Upon completion of this assessment, they will be eligible to participate in the MB-BP training. Individuals in the intervention group will be assessed at 1 year follow up with a subset of measures (see Table 6.1 Schedule of Evaluation) in order to assess long term effects of the intervention.

#### 7. SAFETY ASSESSMENTS

#### 7.1 Expected Risks and Specification of Safety Parameters

*Meditation-related risks:* NCCIH states that meditation is generally safe for healthy people, but that adverse effects have also been reported. <sup>5</sup> Undesirable side effects and risks of meditation have been documented in more than 40 scientific reports [for reviews see <sup>6-8</sup>] and are listed in the Mindfulness-Based Intervention Guidelines. <sup>9,10</sup> More common, less serious side effects that

have been reported by individuals within the context of MBIs or of individuals who are meditating less than an hour per day include: increased depression, anxiety or panic, reexperiencing of traumatic memories, dissociation, executive dysfunction, headaches/body pain and insomnia. 6,11-16 A few case reports of more serious side effects including mania, psychosis, and suicidality have been reported, mostly in the contexts of intensive retreats (>5 hrs/day) or in conjunction with pre-existing psychopathology. The frequency of serious adverse effects in the context of MBIs is estimated to be less than 1%, although adequate estimates are not available. 18

A number of actions have been taken to minimize meditation-related risks at different stages of the study. During the pre-enrollment stage, individuals with severe mental illness are excluded from the study and all risks are clearly communicated in the consent form. During treatment, meditations are relatively short and interspersed with dyads and reflections. Mindfulness homework assigned as part of the intervention is optional and is recommended to not exceed 1 hour per day. Teachers query participants about their experiences with meditation, and provide corrective feedback or modifications when needed. Developing strategies for working with physical and emotional discomfort is an explicit goal of the program. Because not all participants feel comfortable disclosing difficulties in class, an online "safety check-in" questionnaire will query meditation-related risks (see section 6.2.1). Dr. Ellen Flynn, a licensed psychiatrist, will be available to advise on any psychological events that occur, and provide referrals for treatment if needed. Additionally, Dr. Willoughby Britton will provide expert consult on safety monitoring and reporting, including providing DSMP specific training to research staff and investigators.

Psychological distress: Research subjects participating in this study may have feelings of loss of privacy from being contacted about participating in the study, and possible psychological distress caused by questions asked during the in-person and online questionnaires that bring up painful memories or feelings. However, the resulting potential for injury to research subjects is judged to be minimal. We have already contacted and clinically evaluated thousands of participants from other studies such as the New England Family and Women's Health Initiative using similar assessment procedures to this study, with good responses from the participants. With regard to psychological distress from taking part in the MB-BP intervention, given that screening questions will exclude participants with substantial mental illness, and given the NCCIH statement above that "Meditation is considered to be safe for healthy people." we expect that risk of psychological distress will be low. The risk of increased psychological distress from meditation will be clearly outlined in the consent form and participants will be encouraged to consult with both the course instructor and study staff in the case of any increased distress. Dr. Ellen Flynn, a licensed psychiatrist, will be available to advise on any psychological events that occur, and provide referrals for treatment if needed.

Loss of confidentiality: Likelihood: rare. Minimization: Confidentiality will be maintained by using deidentifying data sets. All paper forms and data collection tools, including the informed consent forms, will be kept in a locked filing cabinet in a secure location. All electronic data files containing identifying information will be encrypted with a cloud-based software. Note that although these measures have been taken to protect participants' personal information, complete confidentiality cannot be guaranteed when transmitting information over the internet. All information obtained from participants will be accessible only to research staff.

Injury due to physical activities: It is possible that injuries could be sustained from (1) the gentle mindful movements (yoga), or (2) physical activities that participants engage in as a result of the intervention encouraging exploration of physical activity as a way to reduce blood pressure. (1) Mindful movements: Participants receive a handout during the orientation showing the yoga

poses that will be offered during the course. They are encouraged to explore limits in their body related to movement, but not to go beyond those limits Participants are asked to listen to what their body is telling them more closely than what the mindful movement instructor is telling them. Modifications of poses are available, including for those limited to chairs or wheelchairs. Participants are encouraged to bring the handout of poses to their health care providers if they have any physical limitations, so that the providers can advise on which poses to do, and which to avoid. (2) Physical activities: Participants are encouraged to explore physical activities that promote strength and conditioning as a way to reduce blood pressure. As with the mindful movements, they are encouraged to explore limits in their body related to movement, but not to go beyond those limits. Participants are asked to listen to what their body is telling them more closely than what the mindful movement instructor is telling them. Furthermore, they are encouraged to ask their healthcare provider about advised physical activities if they have any physical limitations.

Risks associated with fMRI: The fMRI study will be conducted using a 3T MR scanner at UMass Medical School, which has been approved for research and clinical studies in children and adults by the FDA. Magnetic resonance (MR) technology does not use X-rays, but instead uses strong magnetic fields and radio waves. Individuals interested in participating in the fMRI study will complete a screening questionnaire to assess eligibility, including asking whether they have devices that can be affected by MRI or conditions (e.g., claustrophobia, body mass greater than 300 lbs.) that prohibit the ability to be scanned. Participants are screened immediately prior to each MRI scan to ensure participant safety. Significant risks also can arise if ferromagnetic materials are brought into the high magnetic field environment of the scanner and immediate vicinity, as they can become hazardous projectiles. These types of items are not permitted in the scanning area. The MR exams are painless, and except for the pulsating sounds, subjects will not be aware that MR scanning is taking place. With proper safety precautions in terms of the avoidance of metal objects, there are no known health risks associated with MRI. The safety of MRI is reflected in the fact that it is used in standard medical practice without the requirement for informed patient consent. Most people experience no ill effects from the magnetic field, but some report claustrophobia, dizziness, mild nausea, headaches, a metallic taste in their mouth, double vision, or a sensation of flashing lights. These symptoms are transient and resolve quickly after the subject exits the scanner. The technologist will be able to hear subjects at all times and subjects are free to end the procedure at any time. In rare cases, a very slight, uncomfortable tingling of the back due to the rapid switching of the magnetic field has been reported during certain types of scans. Subjects are asked to report this immediately so the scan can be changed to avoid this. Although these precautions will avoid all known risks associated with MR, this procedure may involve risks that are currently unknown. The scanner is noisy, but does not harm hearing. For comfort, subjects will be given earplugs to muffle the noise.

Risk of adverse events during the study: It is possible that some patients will have an adverse event during the study, including increased stress or anxiety. Participants with major mental health conditions, such as schizophrenia, history of psychosis, bipolar depression, suicidal ideation, borderline personality disorder, post-traumatic stress disorder, obsessive compulsive disorder, panic attacks, current alcohol or substance abuse, or an eating disorder are ineligible for the study. We expect risk of adverse events to be very low. For further discussion of AE and SAE monitoring and reporting refer to Section 6.2 below.

*Impact statement:* These risks are considered to be minimal and are addressed in the protocol and consent form.

# 7.2 Methods and Timing for Assessing, Recording, and Analyzing Safety Parameters

Safety monitoring will occur continuously throughout the study using both active and passive monitoring methods outlined and discussed in further detail below. All reported AEs, SAEs, and unanticipated problems will be recorded throughout the study using the data collection systems set up and detailed in the Data and Safety Monitoring Plan (DSMP)

The research staff will record all reportable events with start dates occurring any time after informed consent is obtained but no later than the final 1-year assessment. At each study visit, the research staff will inquire about the occurrence of AE/SAEs since the last visit (or time of most recent reporting). Events will be followed for outcome information until resolution or stabilization or until the grant funding ends.

# 7.3 Adverse Events and Serious Adverse Events, Reporting Procedures, and Follow-up

An adverse event (AE) is generally defined as any unfavorable and unintended diagnosis, symptom, sign (including an abnormal laboratory finding), syndrome or disease which either occurs during the study, having been absent at baseline, or if present at baseline, appears to worsen. A serious adverse event (SAE) is generally defined as any untoward medical occurrence that results in death, is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, or is a congenital anomaly.

Per NCCIH safety monitoring requirements, all AEs and SAEs captured and/or observed involving enrolled study participants will be recorded regardless of their relationship to the study intervention. Below we outline possible AEs and SAEs that may occur related to this research study and intervention; present our procedures for capturing and recoding; and detail the protocol for follow up of AEs. For further discussion of the procedures related to safety monitoring and follow up procedures refer to Section 7.4. Safety Monitoring.

Safety Check-ins: All participants enrolled in the study, regardless of treatment allocation, will receive a two-tiered safety monitoring 'check-in' every 2 weeks during the treatment phase of the study; every month during months 3-6 of the follow-up phase; and at the final 1-year time point. The two-tiered system is designed to detect and follow up on AEs that are at least moderate in severity (interfere with ADL), and to minimize staff and participant burden that would otherwise occur if all mild events were queried and documented.

Tier 1 of the safety check-in involves sending all active, enrolled participants an email (or placing a phone call from a research staff member, if no email provided) containing a link to a brief online survey that queries events with moderate or greater levels of severity. Any participant who endorses one or more tier 1 questions will automatically receive a tier 2 survey and follow-up phone call from study staff.

The Tier 2 survey specifically queries the most common meditation-related side effects (e.g. anxiety, depression, dissociation, flashbacks etc.) using patient-reported outcomes measurement information system (PROMIS) or NeuroQol items (or other validated scales if construct is not available), and PROMIS response options (never- very often).

Additionally, the tier 2 survey will ask participants to provide further detail (i.e., date of onset, symptomology, circumstance surrounding the event, relatedness to the intervention, etc.) regarding the AE/SAE reported in the tier 1 survey. Detail provided will be used to guide the tier 2 phone calls made by research study staff.

*Tier 2 Safety Check-in phone call:* Any participant who indicates that he or she experienced an AE or SAE will then receive a follow up call from a trained research staff member. The purpose of the follow up call will be to further document the details of the AE/SAE, assess need for treatment modification, referrals and reporting.

Research staff members conducting the safety monitoring phone interviews will document the details of the AE/SAE using the Adverse Events Form, which will then be included in the participant file as well as in the annual Data Safety Monitoring Reports presented to the DSMB. Reporting procedures for AEs and SAEs related to the study will be followed including reporting all SAEs to the study PI and DSMB committee chair.

#### 7.3.1 Mental Health

Participants assigned to any treatment group may experience mental health or suicidal ideation during the course of their study involvement. All study participants will be monitored for AEs and SAEs by study staff on a monthly basis until the time of their study completion. Additionally, participants will be asked to complete questionnaires about anxiety, depression and suicidal ideation, specifically the Beck Anxiety Inventory and the Center for Epidemiology Study Depression Scale Revised (CESD-R), at each of their in-person assessments, excluding the one year follow up. Dr. Flynn, a licensed psychiatrist with extensive experience evaluating research participants for clinical deterioration or suicidality, will serve as the study clinician.

Beck Anxiety Inventory (BA): If participant scores ≥26 on the Beck Anxiety Inventory, a safety flag will appear notifying the research assistant (RA) administering the assessment. The RA will then implement the MB-BP safety protocol, which is reviewed and approved by the Brown University IRB. Staff are trained on the safety protocol and a hard copy of the protocol is kept in an accessible location in the assessment office at all times.

Depressive Symptomatology: The CESD-R will be administered during the in-person assessment visits, and scores will be reviewed immediately upon completion of the in-person assessments.

- 1. Sadness (dysphoria): Question numbers 2,4, 6
- 2. Loss of Interest (anhedonia): Question numbers 8, 10
- 3. Appetite: Question numbers 1, 18
- 4. Sleep: Question numbers 5, 11, 19
- 5. Thinking / concentration: Question numbers 3, 20
- 6. Guilt (worthlessness): Question numbers 9, 17
- 7. Tired (fatigue): Question numbers 7, 16
- 8. Movement (agitation): Question numbers 12, 13
- 9. Suicidal ideation: Question numbers 14, 15

Participants are considered to meet criteria for major depressive episode if they have anhedonia or dysphoria nearly every day for the past two weeks, plus symptoms in an additional 4 DSM symptom groups noted as occurring nearly every day for the past two weeks. If participants meet criteria for major depressive episode, a safety flag will appear notifying the research

assistant (RA) administering the assessment. The RA will then implement the MB-BP safety protocol, which is reviewed and approved by the Brown University IRB. Staff are trained on the safety protocol and a hard copy of the protocol is kept in an accessible location in the assessment office at all times.

If participants respond having any suicidal ideation (CES-D questions 14 or 15), staff will again be instructed to follow the IRB approved safety protocol.

#### 7.3.2 Physical Health

Possible atrial fibrillation detected during Heartbeat Detection Task: If possible atrial fibrillation is indicated by the Kardia Mobile device during the "Heart Beat Detection Task" a safety flag will appear notifying the research assistant (RA) administering the assessment. The RA will then implement the MB-BP safety protocol.

Out-of-range blood pressure readings: If during an in-person assessment the participants systolic blood pressure (SBP) and/or diastolic blood pressure (DBP) falls outside of the acceptable range outlined in the safety protocol, the RA will be notified and the IRB approved safety protocol will be implemented.

*Injury due to physical activities:* It is possible that injuries could be sustained from (1) the gentle mindful movements (yoga), or (2) physical activities that participants engage in as a result of the intervention encouraging exploration of physical activity as a way to reduce blood pressure.

- (1) Mindful movements: Participants receive a handout during the orientation showing the yoga poses that will be offered during the course. They are encouraged to explore limits in their body related to movement, but not to go beyond those limits Participants are asked to listen to what their body is telling them more closely than what the mindful movement instructor is telling them. Modifications of poses are available, including for those limited to chairs or wheelchairs. Participants are encouraged to bring the handout of poses to their health care providers if they have any physical limitations, so that the providers can advise on which poses to do, and which to avoid.
- (2) Physical activities: Participants are encouraged to explore physical activities that promote strength and conditioning as a way to reduce blood pressure. As with the mindful movements, they are encouraged to explore limits in their body related to movement, but not to go beyond those limits. Participants are asked to listen to what their body is telling them more closely than what the mindful movement instructor is telling them. Furthermore, they are encouraged to ask their healthcare provider about advised physical activities if they have any physical limitations.

Note that adverse events related to physical injuries will be captured during the routine safety check-ins (discussed above).

#### 7.3.3 Other

Participant Initiated (Passive monitoring): Participants are encouraged to contact meditation instructors and/or study staff if any physical or mental health symptoms arise or other study or meditation-related problems occur. Participants may report AEs at any time throughout the study. Events will be evaluated with the Adverse Events Form by study staff.

Attrition: Reasons for attrition are also an important source of AEs, but are rarely assessed adequately, as participants are unlikely to give honest answers if queried directly by study staff. To increase the accuracy of attrition reason reporting, participants will be asked to complete a brief online Participant-initiated dropout reason survey (see Appendix A7).

Investigator-initiated withdrawals: In rare circumstances, a study participant may be withdrawn from the study and/or intervention by the researcher. In this case, the researcher or other study staff should complete the Attrition information form, and describe reasons for attrition. Note, however, that this scenario would be very unusual, and has not happened once in the in the approximately 130 participants who have gone through the MP-BP study to date. Potential reasons for investigator-initiated withdrawal would be MB-BP classroom or assessment disruption in ways that are causing harm or an unsafe environment for other classroom participants, the instructor, or study staff. The screening questionnaire excludes participants with mental health criteria that puts them at higher risk for disruption. We expect this scenario to occur extremely rarely (as evidenced to date), but remains a possibility.

fMRI Study Safety Monitoring: it is possible participants may experience or report an AE or SAE during their involvement with the fMRI Study. Research staff will use the Adverse Events Form and accompanying documents found in the Appendices to document all AE/SAE discovered at the time of involvement in the fMRI imaging study. The logged events will then be communicated to the Coordinating Center, so that they can be included in the participant file as well as in the annual Data and Safety Monitoring Reports presented to the DSMB. Reporting procedures for AEs and SAEs related to the study will be followed including reporting all SAEs to the study PI and DSMB committee chair.

Non-Response to Treatment: The possibility that the treatment will not yield benefit is another possible risk and will be explained during informed consent procedures. Non-responders (identified as minimal change in medical regimen adherence from baseline assessment) will be provided with referrals to other treatment, if desired.

The data collection systems we have set up to monitor and record AEs and SAEs are specifically designed to avoid double capture. Unique participant identifiers, dates and details surrounding events, as well as steps taken to follow up are recorded.

#### 7.4 Safety Monitoring

Oversight of internal monitoring of the participants' safety will be conducted by the local PI, Dr. Eric Loucks. Oversight of the external Data and Safety Monitoring Committee will be conducted by the chair (Dr. Edmondson). The Data and Safety Monitoring Committee will include experts in cardiology (Choudhary), psychology/psychiatry (Edmondson), epidemiology (Choudhary), and biostatistics (Liu).

Entities Conducting Monitoring: The Institutional Review Board (IRBs) at Brown University will review all research procedures, and will provide oversight. Internal monitoring will be done by the Brown University principal investigator (Dr. Loucks) and the Brown University IRB. The Data Safety Monitoring Committee will provide external monitoring, and will meet annually by phone, video conference, or in-person. They will be provided data annually in order to evaluate potential effects of the RCT on major outcomes (e.g. medical regimen adherence). Any serious adverse effects will be immediately reported to the principal investigator (Loucks) and the committee chair.

What is Monitored: Monitoring is done of all procedures to ensure that they conform to the approved protocol; of unforeseen circumstances that might arise and affect safety; of all reports of serious adverse events as defined in US Department of Health and Human Services regulations for the protection of human research subjects 45 CFR Part 46, and the FDA 312.32 (death, life-threatening experience, new or prolonged hospitalization, persistent or significant disability/incapacity); of other significant adverse events (adverse events that lead to drop out by participant or termination by the investigator); of unexpected adverse events resulting from the study; and of expected adverse events.

Monitoring is done of all study inclusion and exclusion criteria. During this clinical trial, we will notify officials, as mandated by law, if a participant reports intention to harm him/herself or others, or reports child abuse or abuse of an elder. Dr. Ellen Flynn, a licensed psychiatrist, will be available to advise on any psychological events that occur, and provide referrals for treatment if needed.

Frequency of Monitoring: All adverse events will be continuously monitored by the PI as they are documented by the study staff in accordance with the protocol (Please see section 7.3). Participants will be given contact information so that they can inform us of events that occur in between study visits. The PI will meet with staff weekly as schedules allow to review participant progress and to check in about the experiences with the experimental procedures, including adverse events. Any adverse events that are observed and/or reported will be reported to Dr. Loucks and the Data Safety Monitoring Committee chair under the proposed timelines in the DSMP. The Investigators and DSMB members will be available to meet outside of the regularly scheduled meetings (scheduled annually), if necessary, due to concerns regarding a particular participant or any problems that may arise for participants. If necessary, they will make appropriate recommendations for changes in protocol, or terminate the study. The Brown University IRB conducts the monitoring at the continuing reviews as scheduled, whenever modification requests are considered, and upon receiving reports of serious adverse events from the PI or anyone else.

Reporting Plan: Any serious adverse events that are observed and/or reported will be immediately reported to Dr. Loucks and the Data Safety Monitoring Committee Chair. Serious adverse events related to the study are then reported to the Brown University IRB and to NIH. Brown University's IRB requires fatalities related to the study be reported within 24 hours. All serious adverse events related to this study will be reported to the Brown University IRB immediately by telephone and by written report within 48 hours of our receipt of information regarding the event. All other adverse events related to the study will be reported at the continuing review. Serious adverse events related to the study will also be reported in writing to the NIH Project Officer within 48 hours of the PI becoming aware. All serious adverse events related to the study will be reported annually in the Progress Report sent to the NIH Project Officer. Data on all AEs and SAEs will be recorded.

Any actions taken by the IRB, other than acceptance of the adverse event report, will be reported to the NIH along with any changes or amendments to the protocol requested by the IRB in response to these reports. Proposed changes or amendments to the protocol in general must be approved in writing by both the Brown University IRB as well as by the funding agency, NCCIH.

#### 8. INTERVENTION DISCONTINUATION

This study will be stopped prior to its completion if: (1) the intervention is associated with adverse effects that call into question the safety of the intervention; (2) difficulty in study recruitment or retention will significantly impact the ability to evaluate the study endpoints; (3) any new information becomes available during the trial that necessitates stopping the trial.

#### 9. STATISTICAL CONSIDERATIONS

#### 9.1 General Design

Analyses will evaluate (1) whether MB-BP influences self-regulation targets, (2) whether the MB-BP-induced changes in self-regulation targets are associated with changes in medical regimen adherence, and (3) whether MB-BP is associated with medical regimen adherence. Analyses will incorporate generalized linear models (GLM) with properly chosen link functions, performed using generalized estimating equations (GEE) with robust standard error estimators. 245,246 This provides an extension of regression analysis to the case of correlated or repeated observations, allows for inclusion of both continuous and discrete dependent variables, and enables modeling of covariance structures when observations are correlated across time. Following "intention-to-treat" principles, analyses will be conducted on all participants in the randomized controlled trial, regardless of intervention completion. Analyses will use GLM with identity links for normally distributed data. The between-groups independent variable in the GEE analysis is intervention condition, with control conditions as distinct referent groups. Categorical variables will be included in GLM/GEE models as indicator variables with one level chosen as referent. Continuous independent variables such as age and baseline blood pressure would be included as linear terms. In addition, we will include assessment time as a linear term and possibly with an additional quadratic term to capture possible non-linear relationship of time with the outcomes. It is conceivable that one would observe a steeper slope in the initial months that would decrease in the pursuing months. Thus, the use of a quadratic term for assessment time would be able to capture these phenomena. To evaluate self-regulation targets as mediators of the effects of MB-BP on medical regimen adherence, mediation analyses described by Valeri and VanderWeele will be employed.<sup>247</sup> Such analyses will allow for potential interactions between the exposure and mediator of interest and account for potential confounders of the exposure-mediator. mediator-outcome, and exposure-outcome relationships using standard regression techniques. These methods estimate total, indirect and direct effect sizes, as well as statistical variance.247

#### 9.2 Sample Size and Randomization

#### **Treatment Assignment Procedures**

Statistical Power:

Utilizing effect sizes and statistical variance from the Stage 1 MB-BP clinical trial showed an increase of MAIA from baseline of mean 22.6 (SD=6.5) to mean 26.3 (SD=6.0) at 6-month follow-up, demonstrating a 3.7 increase in MAIA score (p<0.001). Power analyses using the T statistic and non-centrality parameter, with alpha (two-tailed) set at 0.05 and beta at 0.2, shows with a MAIA increase of 3.7 in MB-BP vs. control, sample size requirements are 46 per group. With DASH diet score increasing from 2.78 (SD=0.61) at baseline to 3.37 (SD=0.81) at 6-month follow-up in the Stage 1 MB-BP study in the 67% of participants with a low DASH score (<5.5), demonstrating a DASH diet score increase of 0.59 (p<0.001). Using an effect size of 0.5, power analyses using the T statistic and non-centrality parameter

suggest that, with alpha (two-tailed) set at 0.05 and beta at 0.2, a sample size of 33 per group will be sufficient.

Using simulations from Fritz and MacKinnon,<sup>248</sup> for 80% power to detect a mediated effect when effect of exposure on mediator, and mediator on outcome, is of small to medium strength (standardized Cohen's d effect sizes of 0.26-0.39 each), based on Sobel first-order test, we will need 90 participants. Given that 67% of Stage 1 participants had DASH diet score <5.5, recruiting a sample size of 160 participants across the UH2 and UH3 phases (Figure 1), this would allow for 107 participants with low DASH diet to be included in primary mediation analyses with DASH diet score as the outcome. Stage 1 effect sizes on DASH diet score were large Cohen's d (d=0.82). Effect sizes on the primary self-regulation outcome was medium (MAIA Cohen's d=0.59). Assuming associations between the MAIA and DASH diet score are in the small to medium range, the study should be adequately powered for mediation analyses. Please note that Stage 1 analyses also demonstrated significant improvements in other health behaviors, including alcohol consumption and physical activity following the MB-BP intervention. Secondary analyses will evaluate impacts of MB-BP on these health behaviors, but are not adequately powered for mediation analyses due to the lower proportion of participants that do not adhere to these behavioral AHA guidelines (i.e. approximately 15% of participants do not comply to AHA alcohol guidelines, and 32% do not adhere to physical activity guidelines in our Stage 1 sample).

The fMRI imaging analyses (n=24 per group) should be adequately powered, based on power calculations shown in the MINDFUL-PC study below and by power calculations outlined in the fMRI study protocol and MOP. To achieve this, we estimate having to enroll up to 60 eligible study participants into the fMRI study.

For fMRI self-regulation neural targets, resting State Functional Connectivity (rs-FC) will be expressed as correlation coefficients, transformed using Fisher's z-transformation for analysis. rs-FC will be obtained at two time points (baseline: T1; post-training: T2) for participants and controls. We will use a mixed effects model with baseline rs-FC as an additional predictor for the change outcome. There are two elements to the hypotheses – the determination of the significance of the change within group and the comparison of the change in the treatment group compared to the control group. For the comparison in change between treatment and control group, with a mixed analysis of variance (within-subjects rs-FC at T1 and T2, and between-subjects according to intervention; sample size, total n = 48, 24/group), we are able to detect an ES of 0.3 between the two treatment groups with 81.3% power (and an ES of .21 with 81.3% power for within-group mindfulness effect; an ES of 0.23 with 87.7% power for an interaction of treatment and time), with two-sided tests at alpha=0.05. Thus is reasonable power to detect small- to moderate-size differences in BOLD.<sup>249</sup>

Our calculations assume drop-out rates will average around 10-15% across each group, with the control group exhibiting the highest rates of withdrawal and loss to follow up. These estimates are based on the Stage 1 and 2a MB-BP trials in the UH2 phase.

Randomization procedure: Please see Section 3 (study design) above.

Blinding protocol: Please see Section 3 (study design) above.

#### 9.3 Definition of Populations

Please see Section 9.1 for Intention-To-Treat analysis approach.

#### 9.4 Interim Analyses and Stopping Rules

Please see Section 8 for stopping rules and related analyses.

#### 9.5 Outcomes

#### 9.5.1 Primary Outcome

Self-Regulation Primary Outcome: Multidimensional Assessment of Interoceptive Awareness (MAIA), a validated measure of body awareness. 222-224 We hypothesize that MB-BP will significantly improve the MAIA in directions of better self-regulation, compared to control.

#### 9.5.2 Secondary Outcomes

Self-regulation outcomes foster triangulation, including further validated measures of interoceptive awareness (Heartbeat Detection Task, 250,251 Interoceptive Awareness fMRI Task 252-254), stress and emotion regulation (Difficulties in Emotion Regulation Scale, 211 Pittsburgh Stress Battery, 255-259 Perceived Stress Scale, 219,220 Beck Anxiety Inventory, 203-209 CESD-R201,202), attention control (Sustained Attention to Response Task, 228-233), self-compassion (Self-Compassion Scale Short Form 121), and self-efficacy (Self control scale and SECD-6 Scale 260-267).

Medical regimen adherence outcome: Diet, assessed utilizing Dietary Approaches to Stop Hypertension (DASH) eating pattern score, <sup>181</sup> measured via diet history food frequency questionnaire. <sup>182</sup> The measure assesses adherence to JNC-7 guidelines DASH eating pattern score (range 0-8). <sup>181,183</sup>

Medical regimen adherence secondary outcomes: (1) Alcohol consumption: Amount and frequency of alcohol consumption, will be assessed via self-report utilizing standard questions from the behavioral Risk Factor Surveillance Survey.<sup>184</sup> AHA/ACC hypertension clinical practice guideline cut-point of healthy alcohol intake is ≤ 2 drinks (e.g. 24 oz. beer, 10 oz. wine, or 3 oz. 80-proof whiskey) per day in men and ≤1 drink per day in women.<sup>10</sup> Medical regimen adherence will be defined as adherence to JNC-7-recommended behavioral and medication treatment of hypertension.<sup>183</sup> (2) Electronically-Measured Antihypertensive Medication Adherence: measured continuously using electronic medication bottle caps (eCAPS, Ottawa, Canada)<sup>185</sup> (3) Body Mass Index: height and weight directly assessed using standard epidemiologic methods, with change evaluated in participants considered overweight or obese (BMI≥25 kg/m²).<sup>186</sup> (4) Physical activity: We will use the International Physical Activity Questionnaire which has undergone substantial validity and reliability testing.<sup>187-189</sup> Adherence to Joint National Commission-7 (JNC-7) guidelines is 30 min aerobic physical activity ≥4 days per week.<sup>183</sup>

#### 9.6 Data Analyses

Please see Section 9.1 for analytic approach.
### 10. DATA COLLECTION AND QUALITY ASSURANCE

### 10.1 Data Collection Forms

Questionnaire data will typically be collected using Qualtrics, LLC (Provo, UT, USA) survey instruments, so that participants can complete questionnaires on their own time at home within the defined assessment windows, using their computers or smart phones. Exceptions to this include the phone screening questionnaire, and the baseline and follow-up questions on depression and anxiety (described in Section 6.2.2) to allow for a safety protocol to be followed if there are high levels of depression, anxiety or suicidal ideation. In the event that participants are uncomfortable or unable to use a computer for tests data will be collected using hard copies of surveys and entered by a trained member of the research staff.

Assessments of blood pressure, height, weight, and medication use are assessed in-person by trained research assistants blinded to treatment allocation.

Confidentiality of Patient Records: The clinical data will be de-identified but linked. Private information such as name, date of birth, and address for recontacting will be kept in a password protected, encrypted database on a different disk than the clinical data held by the Project Coordinator and used for the purposes of contacting participants. The principal investigator will only be given access to identifiable personal information for the purposes of patient safety or monitoring by the NIH, data safety monitoring boards or HIPPA compliance officer approved agents.

## 10.2 Data Management

Data management will be performed by downloading data at minimum every 2 weeks during active data collection periods, and assessing data for missingness and errors. Data will be maintained in password-protected Microsoft Excel Spreadsheets, and then exported using .csv functions for analysis in SAS software.

Please see Section 10.1 for data collection forms description.

### 10.3 Quality Assurance

### 10.3.1 Training

Describe types and mechanisms of training of staff for the study.

Please see **Appendices E and F** for manuals to perform staff training for assessments. Only trained, experienced, culturally competent interviewers will be hired to perform assessments.

### 10.3.2 Quality Control Committee

There is no formal quality control committee.

### 10.3.3 Metrics

Please see Appendices E and F for quality control metrics of blood pressure and anthropometry assessments.

MB-BP Competency and Treatment Fidelity: Treatment fidelity strategies will be performed in accordance with recommendations of the NIH Behavior Change consortium, specifically ensuring treatment fidelity in the following five areas: study design, training providers, delivery of treatment, receipt of treatment and enactment

of treatment skills,<sup>268</sup> as follows. *Study design*: All session durations will be recorded and any deviations from the planned duration will be documented. All class sessions will be taped (as conditions allow). Audiotapes will undergo a quality assessment audit by research technicians, who will review a ten percent randomly selected sample of the recordings. Research staff completing the audit will conduct competency ratings on these tapes using validated adherence scales (MBCT Adherence Scale, where items 1-11 in the scale are for MBSR, MB-BP and MBCT<sup>269</sup>). Data from the audit will be used to provide detailed feedback to treatment providers. We will ensure equivalent dose across conditions, including meditation, yoga and stress reduction training, through tracking the audio recordings. Possible setbacks in implementation of treatment will be addressed, including having a large pool of MBSR and MB-BP instructors in the event that specific instructors no longer teach classes. Instructor attrition will be tracked.

Provider training: MB-BP will be performed by qualified or certified MBSR instructors<sup>191</sup> with formal training in cardiovascular health (e.g. dietician, physician assistant, health and wellness coach, and those with an Associate's or Bachelor's degree in relevant health sciences), and further certification in MB-BP. MB-BP instructor training involves: (1) An initial 40 hour in-person or online videoconference training where the unique elements of MB-BP are introduced. (2) Two half-day inperson training retreats where MB-BP-specific teaching modules are practiced in peer groups, supervised by the senior MB-BP trainer, with peer and trainer feedback. (3) Studying specific evidence-based articles on hypertension etiology, treatment and prevention, as well as articles synthesizing evidence of mindfulness on hypertension and hypertension risk factors. <sup>10,183,192-194</sup> A written exam evaluates knowledge in this area, for which instructors-in-training need to pass. (4) Supervised teaching of MB-BP in non-study participants is done using the Mindfulness-Based Intervention Teacher Assessment Criteria (MBI-TAC), <sup>1,2,195</sup> and an annotated MB-BP Curriculum Guide until adequate quality is established within predefined criteria.

MBSR teacher certification is fairly extensive, and accreditation occurs through the University of Massachusetts Medical School Center for Mindfulness in Medicine, Health Care and Society, detailed elsewhere. Examples of criteria for becoming a certified MBSR teaching include (i) completion of an eight-week MBSR course as a participant, (ii) completion of several multi-day residential training courses in mindfulness based stress reduction practice and teaching, (iii) substantial experience in teaching MBSR, (iv) strong references letters from colleagues and participants who have taken your MBSR courses, (v) completion of several multi-day mindfulness meditation retreats, (vi) have a graduate degree in a field connected to MBSR (e.g. education, psychology, medicine) or demonstration of equivalent understanding through work experience in a related field. There are 89 registered MBSR programs in Massachusetts (60), RI (9) and CT (20) that offer year-round program including the Center for Mindfulness where MBSR originated. Eligible programs must be 8 weeks and the instructors must have completed the MBSR Instructor certification training to participate in the study.

*Delivery of treatment*: We will assess participants' perceptions of provider warmth and credibility using brief measures based on the validated Working Alliance Inventory,<sup>270</sup> and Therapist Empathy Scale<sup>271</sup> at Weeks 4 and 8 of the intervention. Feedback will be provided to the interventionist, and measures of warmth and

credibility will be adjusted for in sensitivity analyses, to evaluate if results differ when these measures are included vs. excluded.

Receipt of treatment and enactment of treatment skills: Adherence to the prescribed MB-BP practices will be monitored through class attendance, practice logs and diaries. Adherence data will be collected weekly during the course of the intervention. Mindfulness will also be measured through the use of the validated Five Facet Mindfulness Questionnaire<sup>218</sup> as well as by asking about at home mindfulness practices post-intervention.

### 10.3.4 Protocol Deviations

Protocol deviations will be reported to the Brown University IRB and NCCIH. A description of the deviations, and any effects on the protection of human subjects will be documented. Investigator(s) will review protocol deviations and determine on a case by case base which data (if any) will be excluded from the final data set.

### 10.3.5 Monitoring

Please see Section 10.3.4. for description of the monitoring approaches.

### 11. PARTICIPANT RIGHTS AND CONFIDENTIALITY

## 11.1 Institutional Review Board (IRB) Review

The protocol, the informed consent document (**Appendix D**), and any subsequent modifications, will be reviewed and approved by the Brown University IRB responsible for oversight of the study.

#### 11.2 Informed Consent Forms

A signed consent form will be obtained from each participant. The consent form will describe the purpose of the study, the procedures to be followed, and the risks and benefits of participation. A signed copy will be offered to each participant and this fact will be documented in the participant's record.

# 11.3 Participant Confidentiality

The clinical data will be de-identified but linked. Private information such as name, date of birth, and address for recontacting will be kept in a password protected, encrypted database on a different disk that the clinical data help by the Project Coordinator. All paper-based records (i.e. signed consent forms) will be kept in a secure physical location (e.g., locked filing cabinet). All computer entry and networking programs will be done using PIDs only. The principal investigator will only be given access to identifiable personal information for the purposes of patient safety or monitoring by the NIH, data safety monitoring boards or HIPPA compliance officer approved agents. Information will not be released without written permission of the participant, except as necessary for monitoring by IRB, the FDA, the NIH, and the OHRP.

## 11.4 Study Discontinuation

The study may be discontinued at any time by the IRB, the NCCIH, the OHRP, the FDA, or other government agencies as part of their duties to ensure that research

participants are protected.

### 12. COMMITTEES

### Data Safety Monitoring Board:

Oversight of internal monitoring of the participants' safety will be conducted by the PI, Dr. Eric Loucks. Investigators on this application have extensive experience with clinical trials for mindfulness-based interventions and cardiovascular health outcomes. Oversight of the external Data and Safety Monitoring Committee will be conducted by the chair, Dr. Donald Edmondson, PhD, who is Assistant Professor of Behavioral Medicine at Columbia University Medical Center. He is a Psychologist, and has extensive research experience in evaluating effects of stress and psychosocial factors on cardiovascular disease outcomes, along with clinical trials methods expertise.

The Data and Safety Monitoring committee will also include a board-certified cardiologist, Dr. Gaurav Choudhary, and a biostatistician, Dr. Tao Liu. Dr. Choudhary, MD, is Associate Professor of Medicine at Brown University. He is a practicing clinical cardiologist with research in epidemiology and cardiology. He will be able to advise on clinical outcomes and any cardiovascular complications arising from the study. Dr. Liu, PhD, is an Associate Professor of Biostatistics at Brown University, experienced in clinical trials. He will receive all preliminary analyses from the primary statistician, and will have access to all data from the study, to evaluate any evidence of serious adverse effects or other concerns.

These individuals are not associated with this research project and thus work independently of the PI. They are also not part of the key personnel involved in this grant. They are qualified to review the patient safety data generated by this study because of their unique expertise in the areas of cardiology, psychology/psychiatry, epidemiology, and biostatistics.

### Entities Conducting Monitoring

The Institutional Review Board (IRBs) at Brown University will review all research procedures, and will provide oversight. Internal monitoring will be done by the principal investigators (Dr. Loucks) and the Brown University IRB. The Data Safety Monitoring Committee will provide external monitoring, and will meet every six months by phone or in-person. During the randomized-controlled trial phases (phase 3 & 4), they will be provided data every six months to evaluate potential effects of the RCT on the primary outcome (i.e. medical regimen adherence). Any serious adverse effects will be immediately reported to the principal investigator (Loucks) and the committee chair (Edmondson).

# 13. PUBLICATION OF RESEARCH FINDINGS

Any presentation, abstract, or manuscript will be made available for review by the sponsor and the NCCIH prior to submission.

### 14. REFERENCES

1. Crane RS, Eames C, Kuyken W, et al. Development and validation of the mindfulness-based interventions - teaching assessment criteria (MBI:TAC). *Assessment*. 2013;20(6):681-688.

- 2. Crane RS, Kuyken W, Williams JM, Hastings RP, Cooper L, Fennell MJ. Competence in Teaching Mindfulness-Based Courses: Concepts, Development and Assessment. *Mindfulness (N Y)*. 2012;3(1):76-84.
- 3. Crane RS, Brewer J, Feldman C, et al. What defines mindfulness-based programs? The warp and the weft. *Psychol Med.* 2017;47(6):990-999.
- 4. Onken LS, Carroll KM, Shoham V, Cuthbert BN, Riddle M. Reenvisioning Clinical Science: Unifying the Discipline to Improve the Public Health. *Clinical psychological science: a journal of the Association for Psychological Science.* 2014;2(1):22-34.
- 5. Tucker KL, Taylor KS, Crawford C, et al. Blood pressure self-monitoring in pregnancy: examining feasibility in a prospective cohort study. *BMC Pregnancy Childbirth*. 2017;17(1):442.
- 6. Cappuccio FP, Kerry SM, Forbes L, Donald A. Blood pressure control by home monitoring: meta-analysis of randomised trials. *Bmj.* 2004;329(7458):145.
- 7. Kernan WN, Viscoli CM, Makuch RW, Brass LM, Horwitz RI. Stratified randomization for clinical trials. *J Clin Epidemiol*. 1999;52(1):19-26.
- 8. Friedman LM, Furberg CD, DeMets DL. *Fundamentals of Clinical Trials.* New York, NY: Springer; 2010.
- 9. Research Randomizer (Version 4.0) [Computer software]. Retrieved on June 22, 2013, from <a href="http://www.randomizer.org/">http://www.randomizer.org/</a> [computer program]. 2013.
- 10. Whelton PK, Carey RM, Aronow WS, et al. 2017
  ACC/AHA/AAPA/ABC/ACPM/AGS/APhA/ASH/ASPC/NMA/PCNA Guideline for the Prevention, Detection, Evaluation, and Management of High Blood Pressure in Adults: Executive Summary: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. *Hypertension*. 2017.
- 11. Santorelli SF, Kabat-Zinn J. MBSR Curriculum Guide and Supporting Materials.

  Mindfulness Based Stress Reduction Professional Training. . Worcester, MA: University of Massachusetts Center for Mindfulness; 2003.
- 12. World Health Report 2002. Reducing risks, promoting healthy life. World Health Organization. Geneva, Switzerland. <a href="http://wwwwhoint/whr/2002">http://wwwwhoint/whr/2002</a>. 2002.
- 13. Institute of Medicine. *Initial National Priorities for Comparative Effectiveness Research.* Washington, D.C.2009.
- 14. Abbott RA, Whear R, Rodgers LR, et al. Effectiveness of mindfulness-based stress reduction and mindfulness based cognitive therapy in vascular disease: A systematic review and meta-analysis of randomised controlled trials. *Journal of psychosomatic research.* 2014;76(5):341-351.
- 15. Segal ZV, Williams JMG, Teasdale JD, Kabat-Zinn J. *Mindfulness-Based Cognitive Therapy for Depression.* New York, NY: The Guildford Press; 2012.
- 16. Bowen S, Witkiewitz K, Clifasefi SL, et al. Relative Efficacy of Mindfulness-Based Relapse Prevention, Standard Relapse Prevention, and Treatment as Usual for Substance Use Disorders: A Randomized Clinical Trial. *JAMA psychiatry*. 2014.
- 17. Kuyken W, Hayes R, Barrett B, et al. Effectiveness and cost-effectiveness of mindfulness-based cognitive therapy compared with maintenance antidepressant treatment in the prevention of depressive relapse or recurrence (PREVENT): a randomised controlled trial. *Lancet.* 2015;386(9988):63-73.
- 18. Fisher ES, Staiger DO, Bynum JPW, Gottlieb DJ. Creating accountable care organizations: the extended hospital medical staff. *Health affairs (Project Hope)*.26(1):w44-57.
- 19. Bodenheimer T. Patient Self-management of Chronic Disease in Primary Care. *Jama*. 2002;288(19):2469-2469.
- 20. Pincus T. Social Conditions and Self-Management Are More Powerful Determinants of Health Than Access to Care. *Annals of internal medicine*. 1998;129(5):406-406.

- 21. Lorig KR, Mazonson PD, Holman HR. Evidence suggesting that health education for self-management in patients with chronic arthritis has sustained health benefits while reducing health care costs. *Arthritis and rheumatism.* 1993;36(4):439-446.
- 22. Williams GC, Rodin GC, Ryan RM, Grolnick WS, Deci EL. Autonomous regulation and long-term medication adherence in adult outpatients. *Health psychology: official journal of the Division of Health Psychology, American Psychological Association.* 1998;17(3):269-276.
- 23. Tucker CM. Self-Regulation Predictors of Medication Adherence Among Ethnically Different Pediatric Patients With Renal Transplants. *Journal of Pediatric Psychology*. 2001;26(8):455-464.
- 24. Horne R, Weinman J. Self-regulation and Self-management in Asthma: Exploring The Role of Illness Perceptions and Treatment Beliefs in Explaining Non-adherence to Preventer Medication. *Psychology & Health*. 2002;17(1):17-32.
- 25. Bandura A. Perceived self-efficacy in the exercise of control over AIDS infection. *Evaluation and Program Planning.* 1990;13(1):9-17.
- 26. Carver CS, Scheier M. Attention and self-regulation: a control-theory approach to human behavior. Springer-Verlag; 1981.
- 27. Carver CS, Scheier MF. *On the Self-Regulation of Behavior*. Cambridge University Press; 2001.
- 28. Vohs KD, Baumeister RF. Handbook of Self-Regulation, Second Edition: Research, Theory, and Applications. 2010:592.
- 29. Bishop SR, Lau M, Shapiro S, et al. Mindfulness: A proposed operational definition. *Clin Psychol-Sci Pr.* 2004;11(3):230-241.
- 30. Hölzel BK, Lazar SW, Gard T, Schuman-Olivier Z, Vago DR, Ott U. How does mindfulness meditation work? Proposing mechanisms of action from a conceptual and neural perspective. *Perspectives on Psychological Science*. 2011;6:537-559.
- 31. Vago DR. Mapping modalities of self-awareness in mindfulness practice: A potential mechanism for clarifying habits of mind. *Annals of the New York Academy of Sciences*. 2014;1307:28-42.
- 32. Kabat-Zinn J. Full Catastrophe Living (Revised Edition): Using the Wisdom of Your Body and Mind to Face Stress, Pain, and Illness. 2013.
- 33. Segal ZV, Williams JMG, Teasdale JD. Mindfulness-Based Cognitive Therapy for Depression (Second Edition). 2013.
- 34. Acceptance and Commitment Therapy and the New Behavior Therapies, 1-29(The Guilford Press 2004).
- 35. Cullen M. Mindfulness-Based Interventions: An Emerging Phenomenon. *Mindfulness*. 2011;2:186-193.
- 36. Hayes SC. Acceptance and commitment therapy, relational frame theory, and the third wave of behavioral and cognitive therapies. *Behavior therapy.* 2004;35:639-665.
- 37. Samuelson M, Carmody J, Kabat-Zinn J, Bratt MA. Mindfulness-Based Stress Reduction in Massachusetts Correctional Facilities. *The Prison Journal*. 2007;2:254-268.
- 38. Sumter MT, Monk-Turner E, Turner C. The benefits of meditation practice in the correctional setting. *Journal of correctional health care : the official journal of the National Commission on Correctional Health Care.* 2009;15(1):47-57; guiz 81.
- 39. Jha AP, Stanley EA, Kiyonaga A, Wong L, Gelfand L. Examining the protective effects of mindfulness training on working memory capacity and affective experience. *Emotion*. 2010;10(1):54-64.
- 40. Stanley EA, Schaldach JM, Kiyonaga A, Jha AP. Mindfulness-based Mind Fitness Training: A Case Study of a High-Stress Predeployment Military Cohort. *Cognitive and Behavioral Practice*. 2011;18(4):566-576.

- 41. Stanley EA, Jha AP. Mind fitness: Improving operational effectiveness and building warrior resilience. *Joint Force Quarterly.* 2009;55:144-151.
- 42. MLERN, Davidson R, Dunne J, et al. Contemplative Practices and Mental Training: Prospects for American Education. *Child Dev Perspect*. 2012;6(2):146-153.
- 43. Kaiser-Greenland S. *The Mindful Child.* New York: Free Press; 2010.
- 44. Greenberg M, Harris A. Nurturing Mindfulness in Children and Youth: Current State of Research. *Child development perspectives*. 2012; 6(2):161–166.
- 45. Meiklejohn J, Phillips C, Freedman M, et al. Integrating Mindfulness Training into K-12 Education: Fostering the Resilience of Teachers and Students. *Mindfulness*. 2012:1-17.
- 46. Shapiro S, Brown K, Astin J. Toward the Integration of Meditation into Higher Education: A Review of Research Evidence. *Teachers College Record.* 2011;113(3): 493-528.
- 47. McCabe Ruff K, Mackenzie ER. The Role of Mindfulness in Healthcare Reform: A Policy Paper. *Explore: The Journal of Science and Healing*. 2009;5(6):313-323.
- 48. Khoury B, Lecomte T, Fortin G, et al. Mindfulness-based therapy: A comprehensive meta-analysis. *Clinical Psychology Review.* 2013;33:763-771.
- 49. Goyal M, Singh S, Sibinga EMS, et al. Meditation programs for psychological stress and well-being: a systematic review and meta-analysis. *JAMA internal medicine*. 2014;174:357-368.
- 50. Olson KL, Emery CF. Mindfulness and weight loss: a systematic review. *Psychosomatic medicine*. 2015;77(1):59-67.
- 51. Rothman AJ. Toward a theory-based analysis of behavioral maintenance. *Health psychology*. 2000;19:64-69.
- 52. Rothman AJ, Baldwin AS, Hertel AW, Fuglestad PT. Self-Regulation and Behavior Change: Disentangling Behavioral Initiation and Behavioral Maintenance. In: Vohs KD, Baumeister RF, eds. *Handbook of Self-Regulation, Second Edition: Research, Theory, and Applications*. New York, NY: Guilford Press; 2011:106-122.
- 53. Muraven M, Baumeister RF. Self-regulation and depletion of limited resources: does self-control resemble a muscle? *Psychological bulletin.* 2000;126(2):247-259.
- 54. Deci EL, Ryan RM. *Intrinsic Motivation and Self-Determination in Human Behavior*. Springer Science & Business Media; 1985.
- 55. Hettema J, Steele J, Miller WR. Motivational interviewing. *Annual review of clinical psychology.* 2005;1:91-111.
- 56. Westra HA, Arkowitz H, Dozois DJA. Adding a motivational interviewing pretreatment to cognitive behavioral therapy for generalized anxiety disorder: a preliminary randomized controlled trial. *Journal of anxiety disorders*. 2009;23(8):1106-1117.
- 57. Vago DR, Silbersweig DA. Self-awareness, self-regulation, and self-transcendence (S-ART): a framework for understanding the neurobiological mechanisms of mindfulness. *Frontiers in Human Neuroscience*. 2012;6:296.
- 58. Fletcher LB, Schoendorff B, Hayes SC. Searching for Mindfulness in the Brain: A Process-Oriented Approach to Examining the Neural Correlates of Mindfulness. *Mindfulness*. 2010;1:41-63.
- 59. Teper R, Inzlicht M. Meditation, mindfulness and executive control: the importance of emotional acceptance and brain-based performance monitoring. *Social cognitive and affective neuroscience*. 2013;8:85-92.
- 60. Teper R, Segal ZV, Inzlicht M. Inside the Mindful Mind: How Mindfulness Enhances Emotion Regulation Through Improvements in Executive Control. *Current Directions in Psychological Science*. 2013;22:449-454.
- 61. Chiesa A, Serretti A, Jakobsen JC. Mindfulness: top-down or bottom-up emotion regulation strategy? *Clinical psychology review.* 2013;33:82-96.
- 62. Marchand WR. Neural mechanisms of mindfulness and meditation: Evidence from neuroimaging studies. *World Journal of Radiology.* 2014;6:471.

- 63. Fan J, Raz A, Posner M. Attentional Mechanisms. In: Aminoff M, Daroff R, eds. *Encyclopedia of Neurological Sciences*. New York: Elsevier; 2003:292-299.
- 64. Fan J, McCandliss BD, Sommer T, Raz A, Posner MI. Testing the efficiency and independence of attentional networks. *Journal of Cognitive Neuroscience*. 2002;14(3):340-347.
- 65. Langner R, Eickhoff SB. Sustaining attention to simple tasks: A meta-analytic review of the neural mechanisms of vigilant attention. *Psychol Bull.* 2013;139(4):870-900.
- 66. Sturm W, Willmes K. On the functional neuroanatomy of intrinsic and phasic alertness. *Neuroimage*. 2001;14(1 Pt 2):S76-84.
- 67. Ridderinkhof KR, van den Wildenberg WP, Segalowitz SJ, Carter CS. Neurocognitive mechanisms of cognitive control: the role of prefrontal cortex in action selection, response inhibition, performance monitoring, and reward-based learning. *Brain Cogn.* 2004;56(2):129-140.
- 68. Rueda MR, Posner MI, Rothbart MK. The development of executive attention: contributions to the emergence of self-regulation. *Dev Neuropsychol.* 2005;28(2):573-594.
- 69. Dillon DG, Pizzagalli DA. Inhibition of Action, Thought, and Emotion: A Selective Neurobiological Review. *Appl Prev Psychol.* 2007;12(3):99-114.
- 70. van Gaal S, Lamme VA, Fahrenfort JJ, Ridderinkhof KR. Dissociable brain mechanisms underlying the conscious and unconscious control of behavior. *J Cogn Neurosci*. 2011;23(1):91-105.
- 71. Schooler JW, Smallwood J, Christoff K, Handy TC, Reichle ED, Sayette MA. Meta-awareness, perceptual decoupling and the wandering mind. *Trends Cogn Sci.* 2011;15(7):319-326.
- 72. Critchley HD, Wiens S, Rotshtein P, Ohman A, Dolan RJ. Neural systems supporting interoceptive awareness. *Nat Neurosci.* 2004;7(2):189-195.
- 73. Vago DR, Pan H, Silbersweig DA, Stern E. Neural Substrates Underlying Modalities of Awareness in Mindfulness Practice. Paper presented at: American Neuropsychiatric Assocation Annual Meeting2013; Boston, MA.
- 74. Valentine E, Sweet P. Meditation and attention: A comparison of the effects of concentrative and mindfulness meditation on sustained attention. *Mental Health, Religion, and culture.* 1999;2(1):59-70.
- 75. Chan D, Woollacott M. Effects of level of meditation experience on attentional focus: is the efficiency of executive or orientation networks improved? *Journal of Alternative and Complementary Medicine*. 2007;13(6):651-657.
- 76. Davidson RJ, Goleman DJ, Schwartz GE. Attentional and affective concomitants of meditation: a cross-sectional study. *Journal of Abnormal Psychology*. 1976;85(2):235-238.
- 77. Slagter HA, Lutz A, Greischar LL, et al. Mental training affects distribution of limited brain resources. *PLoS biology*. 2007;5(6):e138.
- 78. Lazar SW, Bush G, Gollub RL, Fricchione GL, Khalsa G, Benson H. Functional brain mapping of the relaxation response and meditation. *Neuroreport*. 2000;11(7):1581-1585.
- 79. Brefczynski-Lewis JA, Lutz A, Schaefer HS, Levinson DB, Davidson RJ. Neural correlates of attentional expertise in long-term meditation practitioners. *Proc Natl Acad Sci U S A*. 2007;104(27):11483-11488.
- 80. Tang YY, Ma Y, Wang J, et al. Short-term meditation training improves attention and self-regulation. *Proceedings of the National Academy of Science USA*. 2007:104(43):17152-17156.
- 81. Srinivasan N, Baijal S. Concentrative meditation enhances preattentive processing: a mismatch negativity study. *Neuroreport.* 2007;18(16):1709-1712.

- 82. Pagnoni G, Cekic M. Age effects on gray matter volume and attentional performance in Zen meditation. *Neurobiology of Aging*. 2007;28(10):1623-1627.
- 83. Jha AP, Krompinger J, Baime MJ. Mindfulness training modifies subsystems of attention. *Cognitive, Affective, & Behavioral Neuroscience*. 2007;7(2):109-119.
- 84. Bushell WC. New beginnings: evidence that the meditational regimen can lead to optimization of perception, attention, cognition, and other functions. *Ann N Y Acad Sci.* 2009;1172:348-361.
- 85. Lutz A, Slagter HA, Rawlings NB, Francis AD, Greischar LL, Davidson RJ. Mental training enhances attentional stability: neural and behavioral evidence. *The Journal of neuroscience: the official journal of the Society for Neuroscience.* 2009;29(42):13418-13427.
- 86. Wenk-Sormaz H. Meditation can reduce habitual responding. *Advances in Mind-Body Medicine*. 2005;21:33-49.
- 87. Chambers R, Lo BCY, Allen NB. The impact of intensive mindfulness training on attentional control, cognitive style, and affect. *Cognitive Therapy and Research*. 2008;32(3):303-322.
- 88. Gross JJ. The emerging field of emotion regulation: An integrative review. *Review of General Psychology.* 1998;2:271-299.
- 89. Wallis DJ, Hetherington MM. Emotions and eating. Self-reported and experimentally induced changes in food intake under stress. *Appetite*. 2009;52(2):355-362.
- 90. Cosci F. Nicotine dependence and psychological distress: outcomes and clinical implications in smoking cessation. *Psychology Research and Behavior Management*. 2011;4:119-119.
- 91. Elfhag K, Rössner S. Who succeeds in maintaining weight loss? A conceptual review of factors associated with weight loss maintenance and weight regain. *Obesity reviews : an official journal of the International Association for the Study of Obesity.* 2005;6(1):67-85.
- 92. Wing RR, Papandonatos G, Fava JL, et al. Maintaining large weight losses: the role of behavioral and psychological factors. *Journal of consulting and clinical psychology*. 2008;76(6):1015-1021.
- 93. Magai C, Consedine N, Neugut AI, Hershman DL. Common Psychosocial Factors Underlying Breast Cancer Screening And Breast Cancer Treatment Adherence: A Conceptual Review And Synthesis. *Journal of Women's Health*. 2007;16(1):11-23.
- 94. Farb NA, Segal ZV, Mayberg H, et al. Attending to the present: mindfulness meditation reveals distinct neural modes of self-reference. *Social Cognitive and Affective Neuroscience*. 2007;2(4):313-322.
- 95. Taylor VA, Grant J, Daneault V, et al. Impact of mindfulness on the neural responses to emotional pictures in experienced and beginner meditators. *Neuroimage*. 2011.
- 96. Desbordes G, Negi LT, Pace TW, Wallace BA, Raison CL, Schwartz EL. Effects of mindful-attention and compassion meditation training on amygdala response to emotional stimuli in an ordinary, non-meditative state. *Front Hum Neurosci.* 2012;6:292.
- 97. Holzel BK, Carmody J, Evans KC, et al. Stress reduction correlates with structural changes in the amygdala. *Soc Cogn Affect Neurosci.* 2010;5(1):11-17.
- 98. Barnes VA, Treiber FA, Davis H. Impact of Transcendental Meditation on cardiovascular function at rest and during acute stress in adolescents with high normal blood pressure. *Journal of psychosomatic research*. 2001;51(4):597-605.
- 99. Maclean C, Walton K, Wenneberg S, et al. Altered responses of cortisol, GH, TSH and testosterone in acute stress after four months' practice of Transcendental Meditation (TM). *Ann N Y Acad Sci.* 1994:746:381-384.
- 100. Sudsuang R, Chentanez V, Veluvan K. The effect of buddhist meditation on serum cortisol and total protein levels, blood pressure, pulse rate, lung volume and reaction time. *Physiol Behav.* 1991;50:543-548.

- 101. Carlson LE, Speca M, Faris P, Patel KD. One year pre-post intervention follow-up of psychological, immune, endocrine and blood pressure outcomes of mindfulness-based stress reduction (MBSR) in breast and prostate cancer outpatients. *Brain, behavior, and immunity.* 2007;21(8):1038-1049.
- 102. Ortner CMN, Kilner S, Zelazo PD. Mindfulness meditation and emotional interference in a simple cognitive task. *Motivation and Emotion*. 2007; 31: 271-283.
- 103. Tang YY, Ma Y, Wang J, et al. Short-term meditation training improves attention and self-regulation. *Proc Natl Acad Sci U S A.* 2007;104(43):17152-17156.
- 104. Arch JJ, Craske MG. Mechanisms of mindfulness: emotion regulation following a focused breathing induction. *Behaviour research and therapy*. 2006;44(12):1849-1858.
- 105. Erisman SM, Roemer L. A preliminary investigation of the effects of experimentally induced mindfulness on emotional responding to film clips. *Emotion.* 2010;10(1):72-82.
- 106. Goldin PR, Gross JJ. Effects of mindfulness-based stress reduction (MBSR) on emotion regulation in social anxiety disorder. *Emotion*. 2010;10(1):83-91.
- 107. Brewer JA, Sinha R, Chen JA, et al. Mindfulness training and stress reactivity in substance abuse: results from a randomized, controlled stage I pilot study. Substance abuse: official publication of the Association for Medical Education and Research in Substance Abuse. 2009;30(4):306-317.
- 108. Broderick P. Mindfulness and coping with dysphoric mood: Contrasts with rumination and distraction. *Cognitive Therapy and Research*. 2005;29:501-510.
- 109. Campbell-Sills L, Barlow D, Brown T, Hofmann S. Effects of suppression and acceptance on emotional responses of individuals with anxiety and mood disorders. *Behaviour research and therapy.* 2006;44:1251-1263.
- 110. Kuehner C, Huffziger S, Liebsch K. Rumination, distraction and mindful self-focus: effects on mood, dysfunctional attitudes and cortisol stress response. *Psychol Med.* 2009;39(2):219-228.
- 111. Britton WB, Shahar B, Szepsenwol O, Jacobs WJ. Mindfulness-based cognitive therapy improves emotional reactivity to social stress: results from a randomized controlled trial. *Behavior therapy.* 2012;43(2):365-380.
- 112. Holmes DS. Meditation and somatic arousal reduction. *American Psychologist*. 1984;39(1):1-10.
- 113. Britton WB, Haynes PL, Fridel KW, Bootzin RR. Polysomnographic and subjective profiles of sleep continuity before and after mindfulness-based cognitive therapy in partially remitted depression. *Psychosom Med.* 2010;72(6):539-548.
- 114. Creswell JD, Pacilio LE, Lindsay EK, Brown KW. Brief mindfulness meditation training alters psychological and neuroendocrine responses to social evaluative stress. *Psychoneuroendocrinology*. 2014;44:1-12.
- 115. Bandura A. Self-Efficacy: The Exercise of Control. 1997:604.
- 116. Schwarzer R. Self-Efficacy: Thought Control Of Action. 1992.
- 117. Conner, Mark, Norman, Paul. Predicting Health Behaviour. 2005:385.
- 118. The role of self-efficacy in health self-regulation, 137-152(Hogrefe/Huber 2005).
- 119. Neff KD. The development and validation of a scale to measure self-compassion. *Self and Identity*. 2003;2:223-250.
- 120. Neff KD, Kirkpatrick KL, Rude SS. Self-compassion and adaptive psychological functioning. *Journal of Research in Personality*. 2007;41:139-154.
- 121. Neff KD, Vonk R. Self-compassion versus global self-esteem: two different ways of relating to oneself. *J Pers.* 2009;77(1):23-50.
- 122. Adams CE, Leary MR. Promoting Self–Compassionate Attitudes Toward Eating Among Restrictive and Guilty Eaters. *Journal of Social and Clinical Psychology*. 2007;26:1120-1144.

- 123. Who Benefits from Training in Self-Compassionate Self-Regulation? A Study of Smoking Reduction, Journal of Social and Clinical Psychology(2010).
- 124. Magnus CMR, Kowalski KC, McHugh T-LF. The Role of Self-compassion in Women's Self-determined Motives to Exercise and Exercise-related Outcomes. *Self and Identity*. 2010;9:363-382.
- 125. Terry ML, Leary MR. Self-compassion, self-regulation, and health. *Self and Identity*. 2011;10:352-362.
- 126. Nolen-Hoeksema S, Wisco BE, Lyubomirsky S. Rethinking rumination. *Perspectives on Psychological Science*. 2008;3:400-424.
- 127. Smallwood J, Andrews-Hanna J. Not all minds that wander are lost: The importance of a balanced perspective on the mind-wandering state. *Frontiers in Psychology.* 2013;4.
- 128. McMillan RL, Kaufman SB, Singer JL. Ode to positive constructive daydreaming. *Frontiers in Psychology.* 2013;4.
- 129. Killingsworth MA, Gilbert DT. A wandering mind is an unhappy mind. *Science*. 2010;330:932.
- 130. Epel ES, Puterman E, Lin J, Blackburn E, Lazaro A, Mendes WB. Wandering Minds and Aging Cells. *Clinical Psychological Science*. 2012;1:75-83.
- 131. Smallwood J, Fishman DJ, Schooler JW. Counting the cost of an absent mind: mind wandering as an underrecognized influence on educational performance. *Psychonomic Bulletin & Review.* 2007;14:230-236.
- 132. Braboszcz C, Delorme A. Lost in thoughts: Neural markers of low alertness during mind wandering. *NeuroImage*. 2010;54:3040-3047.
- 133. Mooneyham BW, Schooler JW. The costs and benefits of mind-wandering: a review. Canadian journal of experimental psychology = Revue canadienne de psychologie expérimentale. 2013;67:11-18.
- 134. Brewer JA, Worhunsky PD, Gray JR, Tang Y-Y, Weber J, Kober H. Meditation experience is associated with differences in default mode network activity and connectivity. *Proceedings of the National Academy of Sciences of the United States of America*. 2011;108:20254-20259.
- 135. Farb NAS, Segal ZV, Mayberg HS, et al. Attending to the present: mindfulness meditation reveals distinct neural modes of self-reference. *Social Cognitive and Affective Neuroscience*. 2007;2:313-322.
- 136. Craig A. How do you feel? Interoception: the sense of the physiological condition of the body. *Nature Reviews Neuroscience*. 2002;3:655-666.
- 137. *Interoception and emotion: A neuroanatomical perspective*, 06 272-290(Guilford Press 2008).
- 138. Craig A. The sentient self. Brain Structure & Function. 2010;214:563-577.
- 139. Damasio A, Carvalho GB. The nature of feelings: evolutionary and neurobiological origins. *Nature Reviews Neuroscience*. 2013;14:143-152.
- 140. Herbert BM, Pollatos O. The body in the mind: on the relationship between interoception and embodiment. *Topics in Cognitive Science*. 2012;4:692-704.
- 141. Füstös J, Gramann K, Herbert BM, Pollatos O. On the embodiment of emotion regulation: interoceptive awareness facilitates reappraisal. *Social cognitive and affective neuroscience*. 2013;8:911-917.
- 142. Mehling WE, Wrubel J, Daubenmier JJ, et al. Body Awareness: a phenomenological inquiry into the common ground of mind-body therapies. *Philosophy, ethics, and humanities in medicine: PEHM.* 2011;6:6.
- 143. Lutz A, Brefczynski-Lewis J, Johnstone T, Davidson RJ. Regulation of the neural circuitry of emotion by compassion meditation: Effects of meditative expertise. *PloS one*. 2008;3:e1897.

- 144. Lutz A, Greischar LL, Perlman DM, Davidson RJ. BOLD signal in insula is differentially related to cardiac function during compassion meditation in experts vs. novices. *NeuroImage*. 2009;47:1038-1046.
- 145. Lutz A, McFarlin DR, Perlman DM, Salomons TV, Davidson RJ. Altered anterior insula activation during anticipation and experience of painful stimuli in expert meditators. *NeuroImage*. 2013;64:538-546.
- 146. Lamm C, Singer T. The role of anterior insular cortex in social emotions. *Brain Structure & Function*. 2010:579-591.
- 147. Nakata H, Sakamoto K, Kakigi R. Meditation reduces pain-related neural activity in the anterior cingulate cortex, insula, secondary somatosensory cortex, and thalamus. *Frontiers in psychology.* 2014;5:1489.
- 148. Gard T, Hölzel BK, Sack AT, et al. Pain attenuation through mindfulness is associated with decreased cognitive control and increased sensory processing in the brain. *Cerebral Cortex.* 2012;22:2692-2702.
- 149. Allen M, Dietz M, Blair KS, et al. Cognitive-affective neural plasticity following active-controlled mindfulness intervention. *Journal of Neuroscience*. 2012;32:15601-15610.
- 150. Farb NAS, Anderson AK, Mayberg HS, Bean J, McKeon D, Segal ZV. Minding one's emotions: mindfulness training alters the neural expression of sadness. *Emotion*. 2010:10:25-33.
- 151. Farb NAS, Segal ZV, Anderson AK. Attentional modulation of primary interoceptive and exteroceptive cortices. *Cerebral Cortex*. 2013;23:114-126.
- 152. Farb NAS, Segal ZV, Anderson AK. Mindfulness meditation training alters cortical representations of interoceptive attention. *Social cognitive and affective neuroscience*. 2013;8:15-26.
- 153. Luders E, Kurth F, Mayer EA, Toga AW, Narr KL, Gaser C. The unique brain anatomy of meditation practitioners: alterations in cortical gyrification. *Frontiers in Human Neuroscience*. 2012;6:34.
- 154. Lazar SW, Kerr CE, Wasserman RH, et al. Meditation experience is associated with increased cortical thickness. *Neuroreport.* 2005;16:1893-1897.
- 155. Hölzel BK, Ott U, Gard T, et al. Investigation of mindfulness meditation practitioners with voxel-based morphometry. *Social cognitive and affective neuroscience*. 2008;3:55-61.
- 156. Grant JA, Courtemanche J, Rainville P. A non-elaborative mental stance and decoupling of executive and pain-related cortices predicts low pain sensitivity in Zen meditators. *Pain.* 2011;152:150-156.
- 157. Lutz J, Herwig U, Opialla S, et al. Mindfulness and emotion regulation--an fMRI study. Social cognitive and affective neuroscience. 2014;9:776-785.
- 158. Fox KCR, Nijeboer S, Dixon ML, et al. Is meditation associated with altered brain structure? A systematic review and meta-analysis of morphometric neuroimaging in meditation practitioners. *Neuroscience and biobehavioral reviews*. 2014;43C:48-73.
- 159. Zeidan F, Martucci KT, Kraft Ra, Gordon NS, McHaffie JG, Coghill RC. Brain mechanisms supporting the modulation of pain by mindfulness meditation. *Journal of Neuroscience*. 2011;31:5540-5548.
- 160. Brefczynski-Lewis JA, Lutz A, Schaefer HS, Levinson DB, Davidson RJ. Neural correlates of attentional expertise in long-term meditation practitioners. *Proceedings of the National Academy of Sciences of the United States of America*. 2007;104:11483-11488.
- 161. Kabat-Zinn J. An outpatient program in behavioral medicine for chronic pain patients based on the practice of mindfulness meditation: theoretical considerations and preliminary results. *Gen Hosp Psychiatry*. 1982;4(1):33-47.

- 162. Kabat-Zinn J, Massion AO, Kristeller J, et al. Effectiveness of a meditation-based stress reduction program in the treatment of anxiety disorders. *The American journal of psychiatry.* 1992;149(7):936-943.
- 163. Santorelli S, Bonus K, McCallum C, et al. Mindfulness-Based Stress Reduction: Guidelines and Standards of Practice. *Integrative Medicine Mindfulness Program at University of Wisconsin- Madison and the Center for Mindfulness, University of Massachusetts*. 2004.
- 164. MacCoon DG, Imel ZE, Rosenkranz MA, et al. The validation of an active control intervention for Mindfulness Based Stress Reduction (MBSR). *Behaviour research and therapy*. 2012;50(1):3-12.
- 165. Almeida ND, Loucks EB, Kubzansky L, et al. Quality of parental emotional care and calculated risk for coronary heart disease. *Psychosom Med.* 2010;72(2):148-155.
- 166. Everage NJ, Linkletter CD, Gjelsvik A, McGarvey ST, Loucks EB. Implementation of permutation testing to determine clustering of social and behavioral risk factors for coronary heart disease, National Health and Nutrition Examination Survey 2001-2004. *Annals of epidemiology.* 2013;23(7):381-387.
- 167. Liu SY, Buka SL, Kubzansky LD, Kawachi I, Gilman SE, Loucks EB. Sheepskin effects of education in the 10-year Framingham risk of coronary heart disease. *Soc Sci Med.* 2013;80:31-36.
- 168. Loucks EB, Abrahamowicz M, Xiao Y, Lynch JW. Associations of education with 30 year life course blood pressure trajectories: Framingham Offspring Study. *BMC Public Health*. 2011;11:139.
- 169. Loucks EB, Almeida ND, Taylor SE, Matthews KA. Childhood family psychosocial environment and coronary heart disease risk. *Psychosom Med.* 2011;73(7):563-571.
- 170. Loucks EB, Berkman LF, Gruenewald TL, Seeman TE. Social integration is associated with fibrinogen concentration in elderly men. *Psychosom Med.* 2005;67(3):353-358.
- 171. Loucks EB, Berkman LF, Gruenewald TL, Seeman TE. Relation of social integration to inflammatory marker concentrations in men and women 70 to 79 years. *Am J Cardiol.* 2006;97(7):1010-1016.
- 172. Loucks EB, Britton WB, Howe CJ, Eaton CB, Buka SL. Positive associations of dispositional mindfulness with cardiovascular health: The New England Family Study. *Int J Behav Med.* 2014:DOI 10.1007/s12529-12014-19448-12529.
- 173. Loucks EB, Buka SL, Rogers ML, et al. Education and coronary heart disease risk associations may be affected by early-life common prior causes: a propensity matching analysis. *Annals of epidemiology.* 2012;22(4):221-232.
- 174. Loucks EB, Lynch JW, Pilote L, et al. Life-course socioeconomic position and incidence of coronary heart disease: the Framingham Offspring Study. *American journal of epidemiology*. 2009;169(7):829-836.
- 175. Loucks EB, Magnusson KT, Cook S, Rehkopf DH, Ford ES, Berkman LF. Socioeconomic position and the metabolic syndrome in early, middle, and late life: evidence from NHANES 1999-2002. *Annals of epidemiology*. 2007;17(10):782-790.
- 176. Loucks EB, Taylor SE, Polak JF, Wilhelm A, Kalra P, Matthews KA. Childhood family psychosocial environment and carotid intima media thickness: the CARDIA study. *Soc Sci Med.* 2014;104:15-22.
- 177. Senese LC, Almeida ND, Fath AK, Smith BT, Loucks EB. Associations between childhood socioeconomic position and adulthood obesity. *Epidemiol Rev.* 2009;31:21-51.
- 178. Smith BT, Lynch JW, Fox CS, et al. Life-course socioeconomic position and type 2 diabetes mellitus: The Framingham Offspring Study. *American journal of epidemiology*. 2011;173(4):438-447.

- 179. Altunkan S, Iliman N, Altunkan E. Validation of the Omron M6 (HEM-7001-E) upper arm blood pressure measuring device according to the International Protocol in elderly patients. *Blood pressure monitoring*. 2008;13(2):117-122.
- 180. Tucker KL, Sheppard JP, Stevens R, et al. Self-monitoring of blood pressure in hypertension: A systematic review and individual patient data meta-analysis. *PLoS medicine*. 2017;14(9):e1002389.
- 181. Roger VL, Go AS, Lloyd-Jones DM, et al. Heart disease and stroke statistics--2012 update: a report from the American Heart Association. *Circulation*. 2012;125(1):e2-e220.
- 182. Subar AF, Thompson FE, Kipnis V, et al. Comparative validation of the Block, Willett, and National Cancer Institute food frequency questionnaires: the Eating at America's Table Study. *Am J Epidemiol.* 2001;154(12):1089-1099.
- 183. Chobanian AV, Bakris GL, Black HR, et al. Seventh report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure. *Hypertension*. 2003;42(6):1206-1252.
- 184. Centers for Disease Control and Prevention. *Behavioral Risk Factor Surveillance System Survey (BRFSS) Questionnaire*. Atlanta, GA: US Department of Health and Human Services; 2011.
- 185. Information Mediary Corp. eCAP Validation Information. <a href="http://www.informationmediary.com/ecap">http://www.informationmediary.com/ecap</a>. 2018.
- 186. Loucks EB, Gilman SE, Howe CJ, et al. Education and Coronary Heart Disease Risk: Potential Mechanisms Such as Literacy, Perceived Constraints, and Depressive Symptoms. *Health education & behavior : the official publication of the Society for Public Health Education*. 2014.
- 187. Craig CL, Marshall AL, Sjostrom M, et al. International physical activity questionnaire: 12-country reliability and validity. *Med Sci Sports Exerc.* 2003;35(8):1381-1395.
- 188. Lee PH, Macfarlane DJ, Lam TH, Stewart SM. Validity of the International Physical Activity Questionnaire Short Form (IPAQ-SF): a systematic review. *The international journal of behavioral nutrition and physical activity.* 2011;8:115.
- 189. Loucks EB, Britton WB, Howe CJ, Eaton CB, Buka SL. Positive Associations of Dispositional Mindfulness with Cardiovascular Health: the New England Family Study. *Int J Behav Med.* 2015;22(4):540-550.
- 190. University of Massachusetts Medical School. Center for Mindfulness in Medicine HC, and Society. 2013; <a href="http://www.umassmed.edu/cfm/oasis/ataglance/index.aspx">http://www.umassmed.edu/cfm/oasis/indepth/index.aspx</a>. Accessed April 18, 2013, 2013.
- 191. Evans A, Crane R, Cooper L, et al. A Framework for Supervision for Mindfulness-Based Teachers: a Space for Embodied Mutual Inquiry. *Mindfulness (N Y)*. 2015;6(3):572-581.
- 192. Centers for Disease Control and Prevention. High Blood Pressure. Website: <a href="https://www.cdc.gov/bloodpressure/index.htm">https://www.cdc.gov/bloodpressure/index.htm</a>; last accessed on Sept. 29, 2018. 2018.
- 193. American Heart Association. The Facts About High Blood Pressure. Website: <a href="http://www.heart.org/en/health-topics/high-blood-pressure/the-facts-about-high-blood-pressure">http://www.heart.org/en/health-topics/high-blood-pressure/the-facts-about-high-blood-pressure</a>. Last accessed: September 29, 2018. 2017.
- 194. Crane RS, Soulsby JG, Kuyken W, Williams JMG, Eames C. The Bangor, Exeter and Oxford Mindfulness-Based Interventions Teaching Assessment Criteria for assessing the competence and adherence of mindfulness-based class-based teaching within the UK context. *Document in development*. 2011.
- 195. Bernstein DP, Fink L, Handelsman L, et al. Initial reliability and validity of a new retrospective measure of child abuse and neglect. *The American journal of psychiatry*. 1994:151(8):1132-1136.
- 196. Bifulco A, Bernazzani O, Moran PM, Jacobs C. The childhood experience of care and abuse questionnaire (CECA.Q): validation in a community series. *The British journal of clinical psychology*. 2005;44(Pt 4):563-581.

- 197. Bifulco A, Brown GW, Harris TO. Childhood Experience of Care and Abuse (CECA): a retrospective interview measure. *Journal of child psychology and psychiatry, and allied disciplines.* 1994;35(8):1419-1435.
- 198. Bernstein DP, Ahluvalia T, Pogge D, Handelsman L. Validity of the Childhood Trauma Questionnaire in an adolescent psychiatric population. *J Am Acad Child Adolesc Psychiatry*. 1997;36(3):340-348.
- 199. Spinhoven P, Penninx BW, Hickendorff M, van Hemert AM, Bernstein DP, Elzinga BM. Childhood Trauma Questionnaire: factor structure, measurement invariance, and validity across emotional disorders. *Psychol Assess.* 2014;26(3):717-729.
- 200. Merrick MT, Ford DC, Ports KA, Guinn AS. Prevalence of Adverse Childhood Experiences From the 2011-2014 Behavioral Risk Factor Surveillance System in 23 States. *JAMA Pediatr.* 2018;172(11):1038-1044.
- 201. Andresen EM, Malmgren JA, Carter WB, Patrick DL. Screening for depression in well older adults: evaluation of a short form of the CES-D (Center for Epidemiologic Studies Depression Scale). *Am J Prev Med.* 1994;10(2):77-84.
- 202. Van Dam NT, Earleywine M. Validation of the Center for Epidemiologic Studies Depression Scale--Revised (CESD-R): pragmatic depression assessment in the general population. *Psychiatry Res.* 2011;186(1):128-132.
- 203. Beck AT, Epstein N, Brown G, Steer RA. An inventory for measuring clinical anxiety: psychometric properties. *Journal of consulting and clinical psychology.* 1988;56(6):893-897.
- 204. Dobson KS. An analysis of anxiety and depression scales. *J Pers Assess*. 1985;49(5):522-527.
- 205. Enns MW, Cox BJ, Parker JD, Guertin JE. Confirmatory factor analysis of the Beck Anxiety and Depression Inventories in patients with major depression. *J Affect Disord*. 1998;47(1-3):195-200.
- 206. Fydrich T, Dowdall D, Chambless DL. Reliability and validity of the Beck Anxiety Inventory. *J Anxiety Disord*. 1992:6:55-61.
- 207. Osman A, Kopper BA, Barrios FX, Osman JR, Wade T. The Beck Anxiety Inventory: reexamination of factor structure and psychometric properties. *J Clin Psychol*. 1997;53(1):7-14.
- 208. Kohn PM, Kantor L, DeCicco TL, Beck AT. The Beck Anxiety Inventory-Trait (BAIT): a measure of dispositional anxiety not contaminated by dispositional depression. *J Pers Assess*. 2008;90(5):499-506.
- 209. Piotrowski C. The status of the Beck Anxiety Inventory in contemporary research. *Psychol Rep.* 1999;85(1):261-262.
- 210. Pickering TG, Hall JE, Appel LJ, et al. Recommendations for blood pressure measurement in humans and experimental animals: part 1: blood pressure measurement in humans: a statement for professionals from the Subcommittee of Professional and Public Education of the American Heart Association Council on High Blood Pressure Research. *Circulation*. 2005;111(5):697-716.
- 211. Coleman A, Freeman P, Steel S, Shennan A. Validation of the Omron 705IT (HEM-759-E) oscillometric blood pressure monitoring device according to the British Hypertension Society protocol. *Blood pressure monitoring*. 2006;11(1):27-32.
- 212. Behavioral Risk Factor Surveillance System Survey Data. Department of Health and Human Services, Centers for Disease Control and Prevention; 2018. Accessed March 27 2108.
- 213. Buysse DJ, Reynolds CF, 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. *Psychiatry Res.* 1989;28(2):193-213.

- 214. Buysse DJ, Reynolds CF, 3rd, Monk TH, Hoch CC, Yeager AL, Kupfer DJ. Quantification of subjective sleep quality in healthy elderly men and women using the Pittsburgh Sleep Quality Index (PSQI). *Sleep.* 1991;14(4):331-338.
- 215. Gentili A, Weiner DK, Kuchibhatla M, Edinger JD. Test-retest reliability of the Pittsburgh sleep quality index in nursing home residents. *J Am Geriatr Soc.* 1995;43(11):1317-1318.
- 216. Baer RA, Smith GT, Hopkins J, Krietemeyer J, Toney L. Using self-report assessment methods to explore facets of mindfulness. *Assessment*. 2006;13(1):27-45.
- 217. Karlsson J, Persson LO, Sjostrom L, Sullivan M. Psychometric properties and factor structure of the Three-Factor Eating Questionnaire (TFEQ) in obese men and women. Results from the Swedish Obese Subjects (SOS) study. *Int J Obes Relat Metab Disord*. 2000;24(12):1715-1725.
- 218. Cappelleri JC, Bushmakin AG, Gerber RA, et al. Psychometric analysis of the Three-Factor Eating Questionnaire-R21: results from a large diverse sample of obese and non-obese participants. *Int J Obes (Lond)*. 2009;33(6):611-620.
- 219. Roberti JW, Harrington LN, Storch EA. Further psychometric support for the 10-item version of the perceived stress scale. *J Coll Counsel.* 2006;9:135-147.
- 220. Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. *J Health Soc Behav.* 1983;24(4):385-396.
- 221. Gratz KL, Roemer L. Multidimensional assessment of emotion regulation and dysregulation: Development, factor structure, and initial validation of the Difficulties in Emotion Regulation Scale. *J Psychopathol Behav Assess.* 2004(26):41-54.
- 222. Mehling WE, Gopisetty V, Daubenmier J, Price CJ, Hecht FM, Stewart A. Body awareness: construct and self-report measures. *PLoS One.* 2009;4(5):e5614.
- 223. Mehling WE, Price C, Daubenmier JJ, Acree M, Bartmess E, Stewart A. The Multidimensional Assessment of Interoceptive Awareness (MAIA). *PLoS One*. 2012;7(11):e48230.
- 224. Bornemann B, Herbert BM, Mehling WE, Singer T. Differential changes in self-reported aspects of interoceptive awareness through 3 months of contemplative training. *Frontiers in psychology.* 2014;5:1504.
- 225. Brener J, Liu X, Ring C. A method of constant stimuli for examining heartbeat detection: comparison with the Brener-Kluvitse and Whitehead methods. *Psychophysiology*. 1993;30(6):657-665.
- 226. Fresco DM, Moore MT, van Dulmen MH, et al. Initial psychometric properties of the experiences questionnaire: validation of a self-report measure of decentering. *Behavior therapy*. 2007;38(3):234-246.
- 227. Fresco DM, Segal ZV, Buis T, Kennedy S. Relationship of posttreatment decentering and cognitive reactivity to relapse in major depression. *J Consult Clin Psychol.* 2007;75(3):447-455.
- 228. Robertson IH, Manly T, Andrade J, Baddeley BT, Yiend J. 'Oops!': performance correlates of everyday attentional failures in traumatic brain injured and normal subjects. *Neuropsychologia*. 1997;35(6):747-758.
- 229. Molenberghs P, Gillebert CR, Schoofs H, Dupont P, Peeters R, Vandenberghe R. Lesion neuroanatomy of the Sustained Attention to Response task. *Neuropsychologia*. 2009.
- 230. Fassbender C, Murphy K, Foxe JJ, et al. A topography of executive functions and their interactions revealed by functional magnetic resonance imaging. *Brain Res Cogn Brain Res*. 2004;20(2):132-143.
- 231. Morrison AB, Goolsarran M, Rogers SL, Jha AP. Taming a wandering attention: short-form mindfulness training in student cohorts. *Front Hum Neurosci.* 2014;7:897.
- 232. Cheyne JA, Carriere JS, Smilek D. Absent-mindedness: Lapses of conscious awareness and everyday cognitive failures. *Conscious Cogn.* 2006;15(3):578-592.

December 11, 2018

- 233. Mrazek MD, Smallwood J, Schooler JW. Mindfulness and mind-wandering: Finding convergence through opposing constructs. *Emotion*. 2012.
- 234. May J, Andrade J, Kavanagh DJ, et al. The craving experience questionnaire: a brief, theory-based measure of consummatory desire and craving. *Addiction*. 2014;109(5):728-735.
- 235. Cohen S, Mermelstein R, Kamarck T, Hoberman H. Measuring the functional components of social support. In: Sarason IG, Sarason BR, eds. *Social support: Theory, research and application*. The Hague, The Netherlands: Martinus Nijhoff; 1985.
- 236. Russell D, Peplau LA, Cutrona CE. The revised UCLA Loneliness Scale: concurrent and discriminant validity evidence. *J Pers Soc Psychol.* 1980;39(3):472-480.
- 237. Hays RD, Bjorner JB, Revicki DA, Spritzer KL, Cella D. Development of physical and mental health summary scores from the patient-reported outcomes measurement information system (PROMIS) global items. *Qual Life Res.* 2009;18(7):873-880.
- 238. Baumeister RF. Yielding to temptation: Self-control failure, impulsive purchasing, and consumer behavior. *J Consum Res.* 2002;28(4):670-676.
- 239. Tangney JP, Baumeister RF, Boone AL. High self-control predicts good adjustment, less pathology, better grades, and interpersonal success. *J Pers.* 2004;72(2):271-324.
- 240. Connor KM, Davidson JR. Development of a new resilience scale: the Connor-Davidson Resilience Scale (CD-RISC). *Depression and anxiety*. 2003;18(2):76-82.
- 241. Lorig KR, Sobel DS, Ritter PL, Laurent D, Hobbs M. Effect of a self-management program on patients with chronic disease. *Eff Clin Pract.* 2001;4(6):256-262.
- 242. Debski TT, Kamarck TW, Jennings JR, Young LW, Eddy MJ, Zhang YX. A computerized test battery for the assessment of cardiovascular reactivity. *International journal of biomedical computing*. 1991;27(3-4):277-289.
- 243. Koffarnus MN, Bickel WK. A 5-trial adjusting delay discounting task: accurate discount rates in less than one minute. *Experimental and clinical psychopharmacology*. 2014;22(3):222-228.
- 244. National Center for Complementary and Integrative Health (NCCIH). Meditation: An Introduction. Uses of Meditation in the United States.
- http://nccih.nih.gov/health/meditation/overview.htm#meditation. 2014.
- 245. Liang K-Y, Zeger SL. Longitudinal data analysis using generalized linear models. *Biometrika*. 1986;73(1):13-22.
- 246. Zeger SL, Liang K-Y. Longitudinal data analysis for discrete and continuous outcomes. *Biometrics.* 1986;42:121-130.
- 247. Valeri L, Vanderweele TJ. Mediation Analysis Allowing for Exposure-Mediator Interactions and Causal Interpretation: Theoretical Assumptions and Implementation With SAS and SPSS Macros. *Psychological methods*. 2013.
- 248. Fritz MS, Mackinnon DP. Required sample size to detect the mediated effect. *Psychological science*. 2007;18(3):233-239.
- 249. Cohen J. *Statistical power analysis for the behavioral sciences (2nd ed.).* Hillsdale, NJ: Erlbaum; 1988.
- 250. O'Brien WH, Reid GJ, Jones KR. Differences in heartbeat awareness among males with higher and lower levels of systolic blood pressure. *International journal of psychophysiology: official journal of the International Organization of Psychophysiology.* 1998;29(1):53-63.
- 251. Bornemann B, Singer T. Taking time to feel our body: Steady increases in heartbeat perception accuracy and decreases in alexithymia over 9 months of contemplative mental training. *Psychophysiology*. 2016.
- 252. Avery JA, Drevets WC, Moseman SE, Bodurka J, Barcalow JC, Simmons WK. Major depressive disorder is associated with abnormal interoceptive activity and functional connectivity in the insula. *Biological psychiatry*. 2014;76(3):258-266.

- 253. Farb NA, Segal ZV, Anderson AK. Mindfulness meditation training alters cortical representations of interoceptive attention. *Soc Cogn Affect Neurosci.* 2013;8(1):15-26.
- 254. Lezak MD, Howieson DB, Loring DW. *Neuropsychological Assessment.* 4th ed. New York, NY: Oxford University Press; 2004.
- 255. Kamarck TW, Jennings JR, Pogue-Geile M, Manuck SB. A multidimensional measurement model for cardiovascular reactivity: stability and cross-validation in two adult samples. *Health Psychol.* 1994;13(6):471-478.
- 256. Matthews KA, Katholi CR, McCreath H, et al. Blood pressure reactivity to psychological stress predicts hypertension in the CARDIA study. *Circulation*. 2004;110(1):74-78.
- 257. Matthews KA, Woodall KL, Allen MT. Cardiovascular reactivity to stress predicts future blood pressure status. *Hypertension*. 1993;22(4):479-485.
- 258. Steptoe A, Marmot M. Impaired cardiovascular recovery following stress predicts 3-year increases in blood pressure. *J Hypertens*. 2005;23(3):529-536.
- 259. Steptoe A, Kivimaki M. Stress and cardiovascular disease. *Nature reviews Cardiology*. 2012;9(6):360-370.
- 260. Crane MM, Ward DS, Lutes LD, Bowling JM, Tate DF. Theoretical and Behavioral Mediators of a Weight Loss Intervention for Men. *Ann Behav Med.* 2016;50(3):460-470.
- 261. Wingo BC, Desmond Ra Fau Brantley P, Brantley P Fau Appel L, et al. Self-efficacy as a predictor of weight change and behavior change in the PREMIER trial. *Nutr Educ Behav.* 2013;45(1878-2620 (Electronic)):314-321.
- 262. Timmerman GM, Brown A. The effect of a mindful restaurant eating intervention on weight management in women. *Journal of nutrition education and behavior*. 2012;44(1):22-28.
- 263. Burke V, Mansour J Fau Mori TA, Mori Ta Fau Beilin LJ, Beilin Lj Fau Cutt HE, Cutt He Fau Wilson A, Wilson A. Changes in cognitive measures associated with a lifestyle program for treated hypertensives: a randomized controlled trial (ADAPT). 2008(0268-1153 (Print)).
- 264. Cornelio ME, Godin G, Rodrigues RC, de Freitas Agondi R, Alexandre NM, Gallani MC. Effect of a behavioral intervention of the SALdavel program to reduce salt intake among hypertensive women: A randomized controlled pilot study. *Eur J Cardiovasc Nurs*. 2016;15(3):e85-94.
- 265. Irwan AM, Kato M, Kitaoka K, Ueno E, Tsujiguchi H, Shogenji M. Development of the salt-reduction and efficacy-maintenance program in Indonesia. *Nursing & health sciences*. 2016;18(4):519-532.
- 266. Meuleman Y, Hoekstra T, Dekker FW, et al. Sodium Restriction in Patients With CKD: A Randomized Controlled Trial of Self-management Support. *Am J Kidney Dis.* 2017;69(5):576-586.
- 267. Choi SH, Choi-Kwon S. The effects of the DASH diet education program with omega-3 fatty acid supplementation on metabolic syndrome parameters in elderly women with abdominal obesity. *Nutr Res Pract.* 2015;9(2):150-157.
- 268. Bellg AJ, Borrelli B, Resnick B, et al. Enhancing treatment fidelity in health behavior change studies: best practices and recommendations from the NIH Behavior Change Consortium. *Health Psychol.* 2004;23(5):443-451.
- 269. Segal ZV, Teasdale JD, Williams JM, Gemar MC. The Mindfulness-Based Cognitive Therapy Adherence Scale: inter-rater reliability, adherence to protocol and treatment distinctiveness. *Clin Psychol Psychother*. 2002;9:131-138.
- 270. Horvath AO, Greenberg LS. Development and Validation of the Working Alliance Inventory. *J Couns Psychol.* 1989;36(2):223-233.
- 271. Burns DD, Auerbach A. Therapeutic empathy in cognitive-behavioural therapy: does it really make a difference? In: Salkovskis P, ed. *Frontiers of Cognitive Therapy*. New York: Guilford; 1996.

| 272. | Britton W, Shahar B. Mindfulness Skill Acquisition Scale. <i>University of Arizona</i> . 2003. |
|---|---|

# 15. SUPPLEMENTS/APPENDICES

Note that minor modifications may be made to the individual documents listed in the appendices during the course of the study.

Appendix A MB-BP Curriculum Guide

Appendix B MBSR Curriculum Guide

Appendix C MB-BP Phone Screener (verbal consent process)

Appendix D MB-BP Informed Consent

Appendix E Anthropometric Quality Control Manual

Appendix F Blood Pressure Quality Control Manual